# A PHASE 3, RANDOMIZED, OBSERVER-BLINDED, ACTIVE-CONTROLLED TRIAL TO EVALUATE THE IMMUNOGENICITY AND SAFETY OF A RECOMBINANT QUADRIVALENT NANOPARTICLE INFLUENZA VACCINE (QUAD-NIV) WITH MATRIX-M1™ ADJUVANT AGAINST FLUZONE® QUADRIVALENT IN CLINICALLY STABLE ADULTS ≥ 65 YEARS OF AGE

| Investigational Materials: | Hemagglutinin Nanoparticle Influenza Vaccine, Quadrivalent (Quad-NIV), representing the strains recommended for inclusion in quadrivalent vaccines for the 2019 - 2020 northern hemisphere influenza season, ie, A/Brisbane/02/2018 (H1N1) pdm09; A/Kansas/14/2017 (H3N2); B/Maryland/15/2016; B/Phuket/3073/2013; administered with Matrix-M1 Adjuvant |
|---|---|
| Reference Material: | Fluzone® Quadrivalent (Sanofi Pasteur), a United States (US)-licensed seasonal quadrivalent influenza vaccine manufactured for the 2019 - 2020 influenza season. |
| <b>Protocol Number:</b> | qNIV-E-301 |
| Sponsor: | Novavax, Inc. (Novavax) 21 Firstfield Road Gaithersburg, MD 20878 USA |
| Responsible Clinical Operations Manager: | Novavax, Inc. Gaithersburg, MD 20878 Office: Email: |
| Version & Date: | Version 4.0 – 31 October 2019 |
| Prior Version: | Version 3.0 – 03 September 2019<br>Version 2.0 – 02 July 2019<br>Version 1.0 – 21 May 2019 |

#### **CONFIDENTIAL**

The information in this document is considered privileged and confidential by Novavax, Inc. and may not be disclosed to others except to the extent necessary to obtain Institutional Review Board approval and informed consent, or as required by national and local laws. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed.

#### PROTOCOL APPROVAL PAGE

The principal investigator is responsible for ensuring that all trial site personnel, including sub-investigators and other staff members, conduct this trial according to this protocol, Good Clinical Practice (GCP) and International Conference on Harmonisation (ICH) guidelines, the Declaration of Helsinki, and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations during and after trial completion. The principal investigator also agrees not to disclose the information contained in this protocol or any results obtained from this trial without written authorization.

| Investigational Material(s): | Hemagglutinin Nanoparticle Influenza Vaccine, Quadrivalent (Quad-NIV), representing the strains recommended for inclusion in quadrivalent vaccines for the 2019 - 2020 Northern hemisphere influenza season, ie, A/Brisbane/02/2018 (H1N1) pdm09; A/Kansas/14/2017 (H3N2); B/Maryland/15/2016; B/Phuket/3073/2013; administered with Matrix-M1 Adjuvant |
|---|---|
| Reference Material | Fluzone® Quadrivalent (Sanofi Pasteur), a United States (US)-licensed seasonal quadrivalent influenza vaccine manufactured for the 2019 - 2020 influenza season. |
| Protocol: | qNIV-E-301 |
| Date of Issue: | 31 October 2019 |

I have read and approve the protocol specified above and agree on its content:

# Novavax, Inc.

Signed Electronically

| | Date |
|-------------------------------------|------|
| Novavax, Inc. | |
| Signed Electronically | |
| | Date |
| Novavax, Inc. | |
| Clinical Trial Site | |
| Print Name – Principal Investigator | Date |
| Signature | |

# PROTOCOL CHANGE HISTORY


# Protocol Version 4.0, 31 October 2019 (revised from Version 3.0, 03 September 2019)

The following is a summary of the changes made to this protocol.

| <b>Location of Change</b> | Change/Modification in Version 4.0 |
|---|---|
| Section 7.1.2 | The microneutralization assay has been modified to reflect that the assay "will be qualified before use." |
| Section 7.2.1 | Text has been added to clarify that a limited qualification of the cell-mediated immunity assay will be performed prior to its use in clinical testing. |
| Section 10.6.1 | The Day 28 unblinded data review has been clarified to include all primary endpoints (Hemagglutination inhibition antibody responses assayed with egg-propagated virus) testing of associated Day 28 serum samples for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and safety data through Day 28. Data concerning secondary and exploratory endpoints will be included in the unblinded review of Days 0 and 28 as they become available. |

# Protocol Version 3.0, 03 September 2019 (revised from Version 2.0, 02 July 2019)

The following is a summary of the changes made to this protocol.

| <b>Location of Change</b> | Change/Modification in Version 3.0 |
|---|---|
| Protocol Approval Page | signatory has been updated to Novavax, Inc. |
| Synopsis, Section 6.1.5,<br>Appendices 1 and 3 | The Day 28 Study Visit window has been expanded from ± 2 days to ± 4 days. |

# Protocol Version 2.0, 02 July 2019 (revised from Version 1.0, 21 May 2019)

The following is a summary of the changes made to this protocol.

| <b>Location of Change</b> | Change/Modification in Version 2.0 |
|---|---|
| Protocol Approval Page | signatory has been updated to Novavax, Inc. |
| Synopsis, Section 1.9 | Text has been updated to specify that testing for cell-mediated immunity (CMI) responses will be conducted on a subset of approximately 140 subjects from several pre-designated clinical sites (to target approximately 70 evaluable subjects per treatment group) at Days 0, 7, 28, and 182. |

| <b>Location of Change</b> | Change/Modification in Version 2.0 |
|---|---|
| Synopsis, Sections 2.3, 3.2.3 | An additional exploratory objective and endpoint has been added to reflect assessment of CMI responses in a subset of approximately 140 subjects from several pre-designated clinical sites. |
| Synopsis, Section 3.1, 3.3 | "Site" has been added as a stratification factor. |
| Synopsis, Sections 6.1.2, 6.1.4, Appendix 1 | Text has been added to specify additional blood draws on Days 0, 7, 28, and 182 for a subset of approximately 140 subjects from pre-designated clinical sites for the purposes of testing CMI responses. In addition, text has been added to note that all subjects at several pre-designated CMI testing sites will participate in CMI blood sampling and the Informed Consent document at those sites will be adjusted accordingly. |
| Synopsis, Section 10.4.2 | Text has been added to reflect analysis of exploratory CMI response endpoints will be performed on a subset of approximately 140 subjects from several pre-designated clinical sites (70 subjects per treatment arm) and results may be reported as an addendum to the main clinical study report. |
| Section 7, Appendix 3 | The maximum amount of blood drawn has been updated to 168 mL. Most subjects will provide up to 60 mL of blood in the trial. A subset of approximately 140 subjects from several pre-designated clinical sites participating in CMI assessments will provide up to 168 mL. |
| Section 7.2 | Section has been added to describe laboratory assessments of CMI and T Cell responses based on intracellular cytokine staining. |
| General | Minor changes have been made to improve the readability and consistency of the document. |

# **TABLE OF CONTENTS**

| PR | OTOCOL APPROVAL PAGE | 2 |
|-----|------------------------------------------------------------|----|
| PR | OTOCOL CHANGE HISTORY | 3 |
| TA | BLE OF CONTENTS | 5 |
| LIS | T OF TABLES | 8 |
| | OSSARY OF ABBREVIATIONS | |
| | INICAL PROTOCOL SYNOPSIS | |
| 1 | INTRODUCTION | |
| 1.1 | Influenza Virus | |
| 1.1 | Influenza Disease Burden in Older Adults | |
| 1.3 | Licensed Vaccines Against Influenza Virus for Older Adults | |
| 1.4 | Novavax's Nanoparticle Influenza Vaccines | |
| | 1.4.1 Quadrivalent (Quad-NIV) | |
| | 1.4.2 Trivalent (Tri-NIV) | 23 |
| | 1.4.3 Matrix-M1 Adjuvant | 23 |
| 1.5 | Nonclinical Investigations | 24 |
| | 1.5.1 Matrix-M1-adjuvanted Tri-NIV | 24 |
| | 1.5.2 Other Matrix-M1-adjuvanted Vaccines | 25 |
| 1.6 | Clinical Investigations | 25 |
| | 1.6.1 Summary of Phase 2 Trial (qNIV-E-201) with Quad-NIV | 25 |
| | 1.6.1.1 Safety Through Day 28 | 25 |
| | 1.6.1.2 Immunogenicity Through Day 28 | 26 |
| | 1.6.2 Matrix-M-adjuvanted Vaccines | 27 |
| 1.7 | Trial Rationale | 27 |
| 1.8 | Expected Risks from Vaccination with Quad-NIV With or With | |
| 1.9 | M1 AdjuvantRisks Associated with Fluzone Quadrivalent | |
| | _ | |
| 2 | TRIAL OBJECTIVES | |
| 2.1 | Primary Objectives | |
| 2.2 | Secondary Objectives | |
| 2.3 | Exploratory Objectives | |
| 3 | TRIAL OVERVIEW | |
| 3.1 | Design | |
| 3.2 | Trial Endpoints | |
| | 3.2.1 Primary Endpoints | 32 |

| <b>7.1</b> | Serological Assessments of Immunogenicity | 46 |
|---|---|---|
| | .1.1 Hemagglutination Inhibition (HAI) Assay | |
| | 7.1.1.1 Egg-Propagated HAI | |
| | 7.1.1.2 VLP-based HAI | |
| 7 | .1.2 Microneutralization Assay | 47 |
| 7.2 | Assessments of Cell-Mediated Immunity | 47 |
| 7 | .2.1 Assessment of T Cell Responses Based on Intracellular Cytokine Staining | |
| 7.3 | Retention and Use of Archived Specimens | |
| 8 | TRIAL ASSESSMENT OF SAFETY | 49 |
| 8.1 | Adverse Events | 49 |
| 8 | .1.1 Solicited Adverse Events/Subject Diary | 49 |
| 8 | .1.2 Unsolicited Adverse Events | 50 |
| 8 | .1.3 Vital Sign Abnormalities as Adverse Events | 51 |
| 8 | .1.4 Medically-attended Events and Significant New Medical Conditions | |
| 8.2 | Serious Adverse Events | |
| 8.3 | Safety Reporting Requirements and Timelines for SAEs and Certain Other | |
| | Events | <b> 5</b> 3 |
| 8.4 | Severity | |
| 8.5 | Relationship (Causality) | 56 |
| 9 | TRIAL DATA MANAGEMENT | 57 |
| 9.1 | Recording and Collection of Data | 57 |
| 9.2 | Data Quality Assurance | |
| 9.3 | Monitoring | 57 |
| 9.4 | Audit and Inspection | 58 |
| 9.5 | Adherence to and Changes to the Protocol | 58 |
| 9.6 | Retention of Records | 58 |
| 10 | TRIAL STATISTICAL CONSIDERATIONS | 59 |
| 10.1 | Subject Populations | 59 |
| 10.2 | General | 59 |
| 10.3 | Demographics and Protocol Compliance | 59 |
| 10.4 | Analyses Addressing Protocol Objectives | 59 |
| 1 | 0.4.1 Analyses of Primary Objectives | 59 |
| | 10.4.1.1 Immunogenicity | 59 |
| 1 | 0.4.2 Analysis of Secondary and Exploratory Immunogenicity Objectives | 60 |
| 1 | 0.4.3 Analyses Concerning Safety Objectives | 61 |
| 10.5 | Sample Size Considerations. | |
| 10.6 | Plan for Statistical Summarios and Analyses | 61 |

| | ticle Influenza Vaccine, Quadrivalent Confidential<br>x, Inc. Version 4.0 – 31 October 2019 | qNIV-E-301 Protocol<br>Page 8 |
|---|---|---|
| 10.0 | 5.1 Day 28 Unblinded Data Review | 62 |
| 10.0 | | |
| 10.7 | Computer Methods | |
| | IAL LEGAL AND ETHICAL REQUIREMENTS | |
| | Compliance with Regulatory Requirements | |
| | Ethics Committee | |
| 11.3 | Informed Consent | 64 |
| 11.4 | Required Site Documentation | 64 |
| 11.5 | Subject Confidentiality | 65 |
| 11.6 | Disclosure of Information | 65 |
| 12 RF | FERENCES | 66 |
| | NDIX 1 – QNIV-E-301 TRIAL PROCEDURES SCHEDULE | |
| | NDIX 2 – QNIV-E-301 SUBJECT DIARY CARD (DRAFT) | |
| | - | |
| | NDIX 3 – QNIV-E-301 BLOOD DRAW SCHEDULE | |
| APPEN | NDIX 4 – QNIV-E-301 SUBJECT MEASUREMENT TOOL | 72 |
| | LIST OF TABLES | |
| Table 1 | : Trial Design for qNIV-E-301 | 32 |
| Table 2 | : Programmatically-Determined Protocol Deviations | 45 |
| Table 3 | : Listing of Diary Solicited Events | 50 |
| Table 4 | : Adverse Events of Special Interest | 52 |
| Table 5 | : Definition of Severity Grading for Adverse Events | 55 |
| Table 6 | : Severity Grade Definitions for Solicited Gastrointestinal Adver | |
| Table 7 | | |

# **GLOSSARY OF ABBREVIATIONS**

| Abbreviation or Term | Definition |
|----------------------|----------------------------------------------|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANCOVA | Analysis of Covariance |
| APC | Antigen Presenting Cells |
| C | Celsius |
| CBER | Center for Biologics Evaluation and Research |
| CD | Cluster of Differentiation or Compact Disc |
| CDC | Centers for Disease Control and Prevention |
| CI | Confidence Interval |
| CMI | Cell-Mediated Immunity |
| CMO | Chief Medical Officer |
| $CO_2$ | Carbon Dioxide |
| CQA | Clinical Quality Assurance |
| CRA | Clinical Research Associate |
| CRO | Contract Research Organization |
| CSR | Clinical Study Report |
| CTM | Clinical Trial Manager |
| CTMS | Clinical Trial Management System |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| FDA | Food and Drug Administration |
| GBS | Guillain-Barré Syndrome |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |
| GMR | Geometric Mean Ratio |
| GMT | Geometric Mean Titer |
| HA | Hemagglutinin |
| HAI | Hemagglutination Inhibition |
| HD | High-Dose |
| HEENT | Head, Eyes, Ears, Nose, Throat |
| HIV | Human Immunodeficiency Virus |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |

| Abbreviation or Term | Definition |
|----------------------|----------------------------------------------|
| ICH | International Conference on Harmonisation |
| IDMS | Isotope Dilution Mass Spectrometry |
| IgG | Immunoglobulin G |
| IM | Intramuscular |
| IP | Investigational Product |
| IRB | Investigational Review Board |
| ITT | Intent-to-treat |
| IWRS | Interactive Web Randomization System |
| LLOQ | Lower Limit of Quantitation |
| MAE | Medically-attended Event |
| MDCK | Madin Darby Canine Kidney (cells line) |
| MedDRA | Medical Dictionary for Regulatory Activities |
| μg | Microgram |
| mg | Milligram |
| MHC | Major Histocompatibility Complex |
| $\mu L$ | Microliter |
| mL | Milliliter |
| $\mu M$ | Micromolar |
| mM | Millimolar |
| MMP | Methyl-α-D-mannopyranoside |
| MN | Microneutralization |
| NA | Neuraminidase or Not Applicable |
| NI | Non-inferiority |
| NIV | Nanoparticle Influenza Vaccine |
| nm | Nanometer |
| NP | Nucleoprotein |
| NZW | New Zealand White (rabbits) |
| OD | Optical Density |
| PD | Protocol Deviation |
| PBMC | Peripheral Blood Mononuclear Cell |
| PP | Per Protocol |
| PS | Polysorbate |
| PT | Preferred Term |
| qNIV or Quad-NIV | Nanoparticle Influenza Vaccine, Quadrivalent |

| Abbreviation or Term | Definition |
|---|---|
| RBC | Red Blood Cell |
| RSV F | Respiratory Syncytial Virus Fusion |
| SAE | Serious Adverse Event |
| SCR | Seroconversion Rate |
| SD | Standard Deviation |
| Sf | Spodoptera frugiperda |
| SNMC | Significant New Medical Condition |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| SPR | Seroprotection Rate or Surface Plasmon Resonance |
| TCID | Tissue Culture Infective Dose |
| TGS | Toxicity Grading Scale |
| TMAE | Trimethylaminoethyl |
| TMF | Trial Master File |
| tNIV or Tri-NIV | Nanoparticle Influenza Vaccine, Trivalent |
| VLP | Virus-Like Particle |
| VRBPAC | Vaccine and Related Biological Products Advisory<br>Committee |
| WHO | World Health Organization |
| w/v | Weight to Volume |

# **CLINICAL PROTOCOL SYNOPSIS**

| Protocol<br>Number | qNIV-E-301 |
|---|---|
| Title | A Phase 3, Randomized, Observer-blinded, Active-controlled Trial to Evaluate the Immunogenicity and Safety of a Recombinant Quadrivalent Nanoparticle Influenza Vaccine (Quad-NIV) with Matrix-M1 <sup>™</sup> Adjuvant Against Fluzone® Quadrivalent in Clinically Stable Adults ≥ 65 Years of Age. |
| Sponsor and<br>Clinical Phase | Novavax, Inc., 20 Firstfield Road, Gaithersburg, MD 20878<br>Phase 3 |
| Active<br>Treatment | Hemagglutinin Nanoparticle Influenza Vaccine, Quadrivalent (Quad-NIV), representing the strains recommended for inclusion in quadrivalent vaccines for the 2019 - 2020 Northern hemisphere influenza season, ie, A/Brisbane/02/2018 (H1N1) pdm09; A/Kansas/14/2017 (H3N2); B/Maryland/15/2016; B/Phuket/3073/2013 [VRBPAC 2019, WHO 2019]; administered with Matrix-M1 Adjuvant. |
| Reference<br>Materials | Fluzone® Quadrivalent (Sanofi Pasteur), a United States (US)-licensed seasonal quadrivalent influenza vaccine manufactured for the 2010, 2020 influenza season |
| Dosing and<br>Regimen | influenza vaccine manufactured for the 2019 - 2020 influenza season. All subjects will receive an intramuscular (IM) injection on Day 0 of their assigned test article. Injections will contain 240 µg total hemagglutinin (HA) antigen (ie, 60 µg HA of each strain) co-formulated with 75 µg Matrix-M1 adjuvant; or the recommended dose of 2019 - 20 Fluzone Quadrivalent. |
| Purpose and Rationale | Novavax has developed a novel recombinant hemagglutinin (HA) quadrivalent nanoparticle influenza vaccine (Quad-NIV) for the prevention of disease due to influenza virus in adults ≥ 65 years of age, using a recombinant baculovirus and insect cell technology. With a nanoparticle structure, recombinant wild-type sequenced HAs, and use of Matrix-M1 adjuvant, Quad-NIV may offer several important advantages over existing licensed egg-derived seasonal influenza vaccines, including avoidance of antigenic mismatch due to egg-adaptive mutations; and induction of both broadly cross-reactive antibody responses against emerging drift variants of seasonal influenza viruses [Shinde 2018], and potent cross-reactive polyfunctional CD4+ T cells. In a recent Phase 2, dose-finding, formulation-optimizing trial in adults ≥ 65 years of age, multiple formulations of Quad-NIV, containing HA-based antigens representing the 4 influenza strains recommended for inclusion in the 2018 - 2019 Northern hemisphere seasonal influenza vaccine [VRBPAC 2018, WHO 2018] and co-formulated with Matrix-M1 adjuvant, given intramuscularly, induced robust hemagglutination inhibition (HAI) antibody responses against both homologous A/B and drifted H3N2 strains. Three formulations in particular: formulation A (60 μg HA of each strain in-clinic mixed with 50 μg of Matrix-M1); formulation B (60 μg HA of each strain co-formulated with 75 μg of Matrix-M1); and formulation C (60 μg HA of each strain co-formulated with 75 μg of Matrix-M1), induced comparable HAI antibody responses (using both egg-propagated or wild-type-VLP agglutinins as reagents) against all evaluated homologous and drifted H3N2 strains. In addition, all three formulations outperformed Fluzone® High-Dose on HAI antibody responses to all evaluated homologous and drifted H3N2 strains using the wild-type VLP HAI assays, which assessed the binding of vaccine-induced antibodies to HA sequences reflective of circulating viruses not subjected to egg adaptation. The short-term reactogenicity and over |

| | [VDDDAC 2010] WHO 2010], as formulated with 75 up Matrix M1 adjuvent, as segment to a |
|---|---|
| | [VRBPAC 2019, WHO 2019], co-formulated with 75 µg Matrix-M1 adjuvant, as compared to a US-licensed seasonal quadrivalent influenza vaccine comparator, Fluzone Quadrivalent, to generate data to support licensure of Quad-NIV for the prevention of influenza disease in adults ≥ 65 years of age. |
| Primary<br>Objectives | <ul> <li>To demonstrate the non-inferior immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of hemagglutination inhibition (HAI) (assayed with egg-propagated virus) antibody responses to all Quad-NIV homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) at Day 28 post-vaccination.</li> <li>To describe the safety profile of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, and the comparator in clinically stable adults ≥ 65 years of age. The safety profile will include solicited short-term reactogenicity; 28-day all adverse event (AE) profile; 1-year post-injection medically-attended adverse event (MAE), serious adverse event (SAE), and significant new medical condition (SNMC), including immunologically-mediated adverse events of special interest (AESIs).</li> </ul> |
| Secondary<br>Objectives | • To describe the immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, and of a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of HAI (assayed with both egg-propagated virus and wild-type VLP reagents) antibody responses to all Quad-NIV homologous influenza strains (2 influenza A and 2 influenza B strains) and at least 1 antigenically drifted A or B strain in terms of geometric mean titers (GMTs), geometric mean ratio (GMR), seroconversion rate (SCR), seroprotection rate (SPR) and the baseline adjusted ratio of GMTs between treatment arms at Day 28. An additional time-point at Day 182 may be tested by HAI for these outcomes in a subset of subjects in each treatment group. |
| Exploratory<br>Objectives | • To evaluate the superior immunogenicity of 240 μg Quad-NIV co-formulated with 75 μg Matrix-M1 adjuvant, relative to Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of HAI (assayed with both egg-propagated virus and wild-type VLP reagents) antibody responses against all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and 1-2 antigenically-drifted A and/or B strains at Days 0 and 28 post-vaccination. |
| | • To describe the immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, and of a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of microneutralization (MN) responses to vaccine-homologous and/or antigenically-drifted influenza strains at Days 0 and 28 post-vaccination, in terms of GMTs, GMR, SCR, and the baseline adjusted ratio of GMTs between treatment arms at Day 28 post-vaccination. Note: Due to the time-consuming nature of MN testing, this exploratory objective may be completed in a subset of participants in each study treatment group and/or a subset of strains after the initial study HAI data are complete and reported in an addendum. Laboratory staff will remain blinded as to treatment assignments until all projected MN tests are complete. Similarly, an additional time-point at Day 182 may also be tested. |
| | • To describe the quality and amplitude of cell-mediated immune (CMI) responses in healthy adults $\geq 65$ years of age to vaccination with 240 $\mu g$ Quad-NIV co-formulated with 75 $\mu g$ Matrix-M1 adjuvant, as measured by functional T cell responses based on intracellular cytokine analysis. Additional markers of CMI (eg, memory B cells and/or other T cell subsets) may be evaluated depending on availability/recovery of cell volume. Due to the laborious nature of the cellular assays, they will be performed on subjects from a limited number of participating sites and results may be reported as an addendum to the main clinical study report. |
| Primary<br>Endpoints | • Comparative HAI antibody responses (assayed with egg-propagated virus) on Day 28, summarized in terms of the ratio of geometric mean titers (GMTs) AND seroconversion rate |

| | (a ap.) 1100 |
|---|---|
| | <ul> <li>(SCR) difference, between subjects receiving Quad-NIV or Fluzone Quadrivalent for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains). Non-inferiority for each homologous strain will be demonstrated if: <ul> <li>The lower bound of the two-sided 95% CI on the ratio of the GMTs (GMT<sub>QuadNIV</sub>/GMT<sub>Fluzone</sub>) is ≥ 0.67,</li> </ul> </li> <li>AND</li> </ul> |
| | ○ The lower bound of the two-sided 95% CI on the difference between the SCRs $(SCR_{QuadNIV}\text{-}SCR_{Fluzone})$ is $\geq$ -10%. |
| | • Number and percentage (95% CI) of subjects with solicited local and systemic adverse events over the 7 days post-injection (ie, Day 0 through Day 6, inclusive); all adverse events through 28 days post-injection (ie, Day 0 through Day 27, inclusive); and MAEs, SAEs, and SNMCs – including AESIs – through 1 year post-injection. |
| Secondary<br>Endpoints | HAI antibody titers (assayed with both egg-propagated virus and wild-type VLP reagents) at Days 0 and 28 specific for vaccine-homologous A and B strain(s), and antigenically-drifted influenza strains. An additional time-point at Day 182 may also be tested with a subset of subjects. Derived/calculated endpoints based on these data will include: |
| | <ul> <li>GMT – defined as the antilog of the mean of the log-transformed HAI titers, on Days 0 and 28.</li> <li>Geometric mean ratio (GMR) – defined as the ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs (GMR<sub>Post/Pre</sub>) on Day 28.</li> </ul> |
| | <ul> <li>Seroconversion rate (SCR) – defined as proportion of subjects in a given treatment group with either a baseline reciprocal (Day 0) titer of &lt; 10 and a post-vaccination reciprocal</li> </ul> |
| | titer $\geq$ 40, or a baseline reciprocal (Day 0) titer of $\geq$ 10 and a post-vaccination titer $\geq$ 4-fold higher on Day 28. |
| | <ul> <li>Seroprotection rate (SPR) – defined as the proportion of subjects with a reciprocal HAI<br/>titer ≥ 40 on Day 28.</li> </ul> |
| | O Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers). |
| Exploratory<br>Endpoints | <ul> <li>Comparative HAI antibody responses (assayed with both egg-propagated virus and wild-type VLP reagents) on Day 28, summarized in terms of the ratio of geometric mean titers (GMTs) AND seroconversion rate (SCR) difference, between subjects receiving Quad-NIV or Fluzone Quadrivalent for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and 1-2 antigenically-drifted A and/or B strains.</li> <li>Superior immunogenicity for each strain will be demonstrated if: <ul> <li>The lower bound of the two-sided 95% CI on the ratio of the GMTs (GMT<sub>QuadNIV</sub>/GMT<sub>Fluzone</sub>) is greater than 1.5,</li> </ul> </li> </ul> |
| | <ul> <li>The lower bound of the two-sided 95% CI on the difference between the seroconversion<br/>rates (SCR<sub>QuadNIV</sub>- SCR<sub>Fluzone</sub>) is greater than 10%.</li> </ul> |
| | <ul> <li>Microneutralization (MN) responses: Neutralizing antibody titers specific to<br/>vaccine-homologous A and B strain(s) and/or antigenically-drifted influenza strains, at Days 0<br/>and 28 post-vaccination, as measured by a microneutralization assay. An additional time-point<br/>at Day 182 may also be tested. Derived/calculated endpoints based on these data will include:</li> </ul> |
| | <ul> <li>GMT – defined as the antilog of the mean of the log-transformed neutralizing titer for a given treatment group.</li> <li>GMR – defined as the ratio of post-vaccination and pre-vaccination neutralizing GMTs</li> </ul> |
| | <ul> <li>GMR – defined as the ratio of post-vaccination and pre-vaccination neutralizing GMTs within the same treatment group (designated as GMR<sub>Post/Pre</sub>).</li> <li>SCR – defined as proportion of subjects in a given treatment group with either a baseline</li> </ul> |
| | reciprocal titer of < lower limit of quantitation (LLOQ) and a post-vaccination reciprocal |

- titer 4-fold higher than the LLOQ, or a baseline reciprocal titer of  $\geq$  LLOQ and a post-vaccination reciprocal titer  $\geq$  4-fold higher than the baseline titer.
- o Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).
- Counts and/or proportions of Days 0, 7, 28, and 182 peripheral blood effector memory T cell populations that secrete one or more of IL-2, CD40L, IFN-γ, and TNF-α cytokines following *in vitro* restimulation with HA in subjects selected for cellular immune response monitoring. Counts and/or proportions of additional markers of CMI as appropriate.

#### **Trial Design**

This is a Phase 3, randomized, observer-blinded, active-controlled trial to evaluate the immunogenicity and safety of 240  $\mu g$  Quad-NIV co-formulated with 75  $\mu g$  Matrix-M1 Adjuvant against a licensed comparator in clinically stable adults  $\geq 65$  years of age to be conducted in the United States. Approximately 2650 eligible subjects will be enrolled and randomized at a 1:1 ratio into 1 of 2 treatment groups, as shown in the Trial Design table below. The active group (Group A) and the comparator group (Group B) will each consist of approximately 1325 subjects. Both groups will be stratified by site, age (65 to <75 and  $\geq 75$  years), and history of prior year receipt of the 2018-19 influenza vaccine. On Day 0, all subjects will receive a study treatment as indicated in the Trial Design table by intranuscular (IM) injection. Total injection volumes for Quad-NIV will be 0.5 mL. Trial follow-up for each subject will span approximately 1 year from the Day 0 injection. It is anticipated that a percentage of the randomized trial subjects will not complete the trial. Subjects who withdraw or are discontinued will not be replaced.

#### Trial Design for qNIV-E-301

| | | Day 0 Trial Treatme | ent Injection | | | Subjects Per Group |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Vaccine | HA Dose per Strain,<br>μg<br>(H1N1/H3N2/B <sub>V</sub> /B <sub>Y</sub> ) | Matrix-M1<br>Adjuvant<br>Dose | Injection<br>Volume | Treatment Arm | |
| A | Quad-NIV | 60, 60, 60, 60 | 75 µg | 0.5 mL | Non-dominant | 1325 |
| В | | 2019-20 Fluzone Qu | ıadrivalent <sup>[1]</sup> | | TVOII-dominant | 1325 |
| | | | • | | Total Trial Subjects | 2650 |

Abbreviations:  $B_y = B$  Victoria lineage;  $B_Y = B$  Yamagata lineage; HA = Hemagglutinin

Note: All subjects will receive a single vaccination by IM injection in their non-dominant arm on Day 0. If the non-dominant arm is not available for injection, then the dominant arm will be used.

#### Trial Visit Procedures

All subjects will undergo procedures summarized in the Schedule of Events table and described in detail below.

#### Day 0 - Screening Visit

Clinically stable male and female volunteers, ≥ 65 years of age, who have provided written informed consent to participate in the trial and who are able to comply with trial requirements, will have the following procedures performed: review of inclusion and exclusion criteria; medical history, including influenza vaccination history during the previous 3 years (with emphasis on the 2018-19 vaccine) and history of adverse reactions to prior influenza vaccines and allergies; medication history; physical examination of HEENT (head, eyes, ears, nose, and throat), abdomen, extremities, and at least inguinal, cervical, and axillary nodes, gross motor function, and skin; vital signs (heart rate, blood pressure, respiratory rate, and oral temperature), height, and weight; and assessment of concomitant medications. Note that further procedures may be performed at the investigator's discretion in order to adequately screen subjects against eligibility criteria. Potential subjects who meet all inclusion criteria and none of the exclusion criteria (see Inclusion / Exclusion Criteria ) may be enrolled. Note: Subjects should be free of acute illness (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature  $\geq 38.0^{\circ}\text{C}$ ) in order to receive the test article injection. Subjects presenting with an acute illness on screening may return to the trial site within the next 7 days, provided the enrollment timelines allow, to receive their injection provided symptoms have resolved.

#### Day 0 - Trial Treatment Injection Visit

<sup>[1]</sup> Fluzone Quadrivalent will be administered at the manufacturer's recommended dose and volume.

All subjects who have eligibility confirmed will have blood drawn for baseline immunogenicity testing (eg, HAI and MN titers; 20 mL), and then be randomized to 1 of 2 treatment groups.


A subset of approximately 140 subjects from several pre-designated clinical sites (to target approximately 70 evaluable subjects per treatment group) will provide additional blood samples (27 mL per visit) at 4 time points (ie, Days 0,7, 28, and 182) to support testing of cell-mediated immune responses (CMI). Note: All subjects at several pre-designated CMI testing sites will participate in CMI blood sampling and the Informed Consent document at those sites will be adjusted accordingly.

Subjects will then receive a single IM injection of their assigned treatment into the deltoid muscle of the non-dominant arm. (If the non-dominant arm is not available due to post-surgical changes, skin changes, or prior injury, the dominant arm may be used). Subjects will be monitored in the clinic for approximately 30 to 60 minutes following injection with trial treatment for the occurrence of any local injection site or systemic reactions, including evaluation of vital signs.

Starting on vaccination day (Day 0) and for 6 days thereafter (Day 0 through Day 6 inclusive), subjects will maintain diaries for daily recording of their body temperature and any adverse event spontaneously experienced. In addition, the following local injection site and systemic reactions will be solicited by diary: injection site (local) events - pain, bruising, redness, and swelling; general systemic events - oral temperature, chills, muscle pain, joint pain, diarrhea, nausea, vomiting, headache, and fatigue; and facial/respiratory systemic events - cough, difficulty breathing, difficulty swallowing, hoarseness, chest tightness, sore throat, wheezing, eye redness, and facial swelling. Subjects will also be asked to record any concomitant medications, physician visits, or hospitalizations associated with these solicited adverse events.

#### Follow-up Telephone Contacts and In-clinic Visits

Safety follow-up visits will be performed by scripted telephone contact on Day 3 ( $\pm$  1 day) to query for any Grade 3 solicited or unsolicited event and/or SAE experienced and concomitant medications taken for these events since the last visit. Subjects who report a Grade 3 event and/or SAE may be asked to return to the clinic for an unscheduled visit at the investigator's discretion.

On Days 7, 28, and 182, a subset of approximately 140 subjects who were enrolled at several pre-designated clinical sites, and who provided blood for CMI responses at Day 0, will provide additional blood samples for post-vaccination CMI responses (27 mL per visit).

On Day 28 (± 4 days), all subjects will return to the clinic for collection of vital signs, diary review, to provide blood samples for post-vaccination immunogenicity testing (20 mL), and to report any AEs, MAEs, SNMCs, and SAEs occurring since the last visit, and any concomitant medications taken. Subjects will return to the clinic again on Day 182 (± 7 days) for collection of vital signs, to provide blood samples for post-vaccination immunogenicity testing (20 mL), and to report any MAEs, SNMCs, and SAEs occurring since the last trial visit, and any concomitant medications taken for these events.

Additional safety telephone contacts will occur on Days 90 (± 7 days) and 364 (± 14 days) to query for any MAEs, SNMCs, and SAEs occurring since the last trial visit, and any concomitant medications taken for these events.

#### **Schedule of Events:**

| Trial Day: | 0 | 3 | 7 | 28 | 90 | 182 | 364 |
|---|---|---|---|---|---|---|---|
| Window (days): | | ± 1 | ± 1 | ± 4 | ± 7 | ± 7 | ± 14 |
| Trial Procedures | | | | | | | |
| Trial Informed Consent | X | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | |
| Medical/Medication<br>History | X | | | | | | |
| Physical Exam | X | | X [4] | X [4] | | X [4] | |
| Vital Signs | X [1] | | X | X | | X | · |

| | | 37 | | 1 | 37 | | 37 | |
|---|---|---|---|---|---|---|---|---|
| | Serology | X<br>X <sup>[5]</sup> | | X <sup>[5]</sup> | X<br>X <sup>[5]</sup> | | X<br>X <sup>[5]</sup> | |
| | PBMC for CMI | l | | X <sup>[3]</sup> | X <sup>[3]</sup> | | X <sup>[3]</sup> | |
| | Trial Treatment Injection | X | 37 | 37 | 37 | 37 | 37 | 77 |
| | Adverse Event Review [2] | X | X | X | X | X | X | X |
| | Concomitant Medications<br>Review [2] | X | X | X | X | X | X | X |
| | Subject Diary Review | | | | X [3] | | | |
| | End of Trial | | | | | | | X |
| | Note: Procedures shaded in grey are | | | | | | | |
| | [1] Vital signs to be captured pre-vaccination and between 30 to 60 minutes post-vaccination. [2] All adverse events and concomitant medications taken will be collected through Day 28; thereafter, only MAEs, SAEs, and SNMCs and medications taken for these events will be collected. [3] The subject diary will be reviewed by the investigator and collected at the Day 28 visit. [4] If needed, a physical examination may be performed, based on the investigator's discretion. [5] To be collected from a subset of approximately 140 subjects from several pre-designated clinical sites. | | | | | | | |
| Inclusion | Subjects must meet the follow | _ | | | _ | | | |
| Criteria | Clinically-stable adult m | | | • | _ | | • | 1 or more |
| | chronic medical diagnose | | | • | | • | | |
| | Ambulatory status, | | | | | | residenti | al facility |
| | providing minimal as • Absence of changes i | | | | | | + fail | m tovioitu |
| | <ul><li>Absence of changes i</li><li>Absence of medical e</li></ul> | | | | | | | - |
| | and | vents qua | mymg as | scrious ac | iverse eve | iits witiiii | the prior | 2 monuis, |
| | Absence of known | , current, | and life | -limiting | diagnose | s which | render su | ırvival to |
| | completion of the pro | | | | | | | |
| | 2) Willing and able to give | informed | consent p | rior to tria | ıl enrollm | ent, and | | |
| | 3) Living in the community and able to attend trial visits, comply with trial requirements, and | | | | | | | |
| | provide timely, reliable, | | | | | • | | |
| Exclusion | Subjects will be excluded if the | • | • | _ | | | | |
| Criteria | Participation in research 45 days before planned d | ate of stud | ly vaccina | ition. | | | gic / devid | ce) within |
| | 2) Participation in any previ | ous Nova | vax influe | nza vacci | ne clinica | l trial(s). | | |
| | 3) History of a serious react Fluzone Quadrivalent or | | | za vaccina | ation, kno | wn allerg | y to const | tituents of |
| | _ | | | within 6 | waalsa fa | llowing a | provious | influenza |
| | 4) History of Guillain-Barro vaccine. | | | | | | | |
| | 5) Received any vaccine in t within 6 months preceding | | | | l vaccinati | ion and an | y influenz | za vaccine |
| | 6) Any known or suspected in history and/or physical expected in the suspect of t | | | illness, co | ongenital | or acquire | d, based o | n medical |
| | 7) Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. | | | | | | | |
| | An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of | | | | | | | |
| | prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted. | | | | | | | |
| | 8) Administration of immun the administration of the | | | ny blood p | products v | vithin the | 3 months | preceding |
| | 9) Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration). | | | | | | | |
| | 10) Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results | | | | | | | |

| (including neurologic or psychiatric conditions deemed likely to impair the quality of safety |
|---|
| reporting). |

- 11) Known disturbance of coagulation.
- 12) Suspicion or recent history (within 1 year of planned vaccination) of alcohol or other substance abuse.

#### Statistical Methods

#### General

Continuous variables will be presented by summary statistics (eg, mean and standard deviation [SD] for the non-immunogenicity endpoints; geometric means and their 95% CI for the immunogenicity endpoints). Categorical variables will be presented by frequency distributions (frequency counts and percentages for the non-immunogenicity endpoints; percentages and their 95% CIs for the immunogenicity endpoints).

#### **Analyses Concerning the Primary Immunogenicity Objective**

The per-protocol (PP) population (ie, randomized subjects who received the assigned dose of the test article according to the protocol, have HAI serology results at Day 0 and Day 28, and have no major protocol deviations) will be the primary population for immunogenicity analysis. A separate intent-to-treat (ITT) population analysis will not be produced unless > 5% of at least 1 treatment group is excluded from the PP population. No missing data will be imputed. For GMTs and GMRs, titers reported below the lower limit of quantitation (LLOQ, ie, below the starting dilution of assay reported as "< 10") will be set to half that limit (ie, 10/2 = 5).

For purposes of determining non-inferiority (and exploratory superiority) in immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, for all Quad-NIV homologous influenza strains (2 influenza A and 2 influenza B strains) at 28 days post-vaccination, derived/calculated endpoints will include:

- Two-sided 95% CIs for the ratio of Day 28 post-vaccination GMTs between Quad-NIV and Fluzone Quadrivalent will be constructed using log normal distribution. The log<sub>10</sub> values will be used to construct a CI using the analysis of covariance (ANCOVA) with treatment group and baseline at Day 0 (adjusted for intergroup variation in baseline [pre-vaccination] titers) as the covariates under two-sided type I error rate of 0.05. No type I error rate adjustments will be made. The mean difference and the corresponding CI limits will then be exponentiated to obtain the ratio of GMT and the corresponding CI.
- Two-sided 95% CIs for the difference of the SCRs between Quad-NIV and Fluzone Quadrivalent will be based on the Newcombe hybrid score (METHOD = SCORE riskdiff-option for PROC FREQ in SAS).

#### Analyses Concerning the Secondary and Exploratory Immunogenicity Objectives

Immunogenicity of 240  $\mu g$  Quad-NIV co-formulated with 75  $\mu g$  Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, based on HAIs (assayed with both egg-propagated virus and wild-type VLP reagents) for all vaccine-homologous influenza A and B strains, and at least 1 antigenically-drifted A or B strain at Day 28 post-vaccination, will be measured in terms of:

- GMT defined as the antilog of the mean of the log-transformed HAI titers, on Days 0 and 28.
- Geometric mean ratio (GMR) defined as the ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs (GMR<sub>Post/Pre</sub>) on Day 28.
- Seroconversion rate (SCR) defined as proportion of subjects in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40,

- or a baseline reciprocal (Day 0) titer of  $\geq$  10 and a post-vaccination titer  $\geq$  4-fold higher on Day 28.
- Seroprotection rate (SPR) defined as the proportion of subjects with a reciprocal HAI titer
   ≥ 40 on Day 28.
- Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).

An additional time-point at Day 182 may also be tested.

Microneutralization (MN) responses at Days 0 and 28 post-vaccination will include:

- GMT defined as the antilog of the mean of the log-transformed neutralizing titer for a given treatment group.
- GMR defined as the ratio of post-vaccination and pre-vaccination neutralizing GMTs within the same treatment group (designated as GMR<sub>Post/Pre</sub>).
- SCR defined as proportion of subjects in a given treatment group with either a baseline reciprocal titer of < lower limit of quantitation (LLOQ) and a post-vaccination reciprocal titer 4-fold higher than the LLOQ, or a baseline reciprocal titer of ≥ LLOQ and a post-vaccination reciprocal titer ≥ 4-fold higher than the baseline titer.
- Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).

An additional time-point at Day 182 may also be tested.

Analysis of exploratory CMI response endpoints will be performed on a subset of approximately 140 subjects from several pre-designated clinical sites (70 subjects per treatment arm) and results may be reported as an addendum to the main clinical study report.

#### **Analyses Concerning Safety Objectives**

Safety analysis will be descriptive and based on the safety population, defined as all subjects who received a dose of trial treatment, analyzed as actually treated. Safety will be summarized overall and by individual treatment arms based on solicited short-term reactogenicity post-injection on Day 0 - 6, 28-day all AE profile by MedDRA preferred term, and 1-year MAE, SAE, and SNMC profiles post-injection on Day 0. All AEs, including MAEs, SAEs, and SNMCs, will be tabulated by severity, related (possibly, probably, or definitely vs non-related per investigator assessment), and severe and related. The number and percentage (with 95% CI) of subjects in each treatment group with a given term will be summarized. A listing and narratives of SAEs will also be produced.

#### Sample Size Considerations

This study has a single comparison between Quad-NIV and Fluzone Quadrivalent at Day 28 post-vaccination for the primary immunogenicity objective. No adjustment of the Type I error rate for multiple comparisons is warranted since the simultaneous successes of all 8 comparisons planned for the 4 strains contained in the vaccines and the two endpoints (GMT and SCR) are required for the demonstration of the primary non-inferiority objective of the study.

Non-inferiority is defined as the lower bound of the 2-sided 95% CI on the ratio of GMTs (Quad-NIV vs Fluzone)  $\geq$  0.67 (ie, unadjusted 1-sided p-value < 0.025 against the null hypothesis of H<sub>0</sub>: Ratio of GMT < 0.67) and the lower bound of the two-sided 95% CI on the difference of the SCRs (Quad-NIV - Fluzone)  $\geq$  -10% (ie, unadjusted 1-sided p-value < 0.025 against the null hypothesis of H<sub>0</sub>: Difference of SCRs < -10%).

For the calculation of sample size estimation, we used assumptions of true differences, ie, the ratio of GMTs (Quad-NIV vs Fluzone Quadrivalent) is 1.0 for all 4 homologous strains, and the difference of the SCRs is -2% for each of the 4 homologous strains, based on the average performance in the previous trial (qNIV-E-201). To achieve an overall 90% power (ie, ~ 97.5% power for each of the 4 strains) to demonstrate a non-inferiority margin for SCR difference of -10%, the SCR of the reference group (Fluzone Quadrivalent) is assumed to be 0.5 and the SCR of treatment group (Quad-NIV) is assumed to be 0.48 under the null hypothesis of inferiority (H<sub>0</sub>: Difference of SCRs < -10%). The significance level of the testing is 0.025. Sample size was estimated to be 1195 in each group by assuming equal size in each group. The sample size accounted for a 10% attrition rate for the per-protocol population such that the primary analysis

population for all immunogenicity endpoints will be 1325 in each group.

In a previous trial (qNIV-E-201), the observed vaccine-homologous strain-specific standard deviations of  $\log_{10}$  HAI titers ranged from approximately 0.3 (B/Colorado/06/2017 and B/Phuket/3073/2013) to approximately 0.4 (A/Singapore/INFIMH-16-0019/2016 and A/Michigan/45/2015). The calculated power for each strain, unadjusted for multiple comparisons, is close to 100% to detect a 1.5-fold difference in GMTs. For 4 strains, this study is designed to exclude a GMT ratio of < 0.67 with 100% power. Therefore, for demonstrating non-inferiority for 4 strains with the true ratio of GMTs of 1.0 and the true SCR differences of -2%, this study provides  $\geq$  90% overall power.

For safety endpoints, the probability of observing at least 1 adverse event among 1325 subjects for Quad-NIV is > 90% if the true rate of such events is 0.18%. With 1325 subjects for Quad-NIV, observing no adverse events of interest (eg, vaccine-related SAE) would represent an upper bound of the 1-sided 95% CI on the percentage of such event is 0.2%.

#### 1 INTRODUCTION

# 1.1 Influenza Virus

Influenza is an airborne, respiratory pathogen that is generally transmitted by inhalation of infectious droplets of respiratory secretions, although transmission via fomites can also occur. Infections in humans often lead to annual outbreaks and worldwide epidemics, mainly in the winter seasons. The virus infects the upper respiratory epithelium of the nose, throat, bronchi, and occasionally the lungs. Clinical characteristics of influenza infection include sudden onset of fever, myalgia, headache, severe malaise, dry cough, sore throat, and rhinitis. Although the majority of people recover within 1 to 2 weeks without any major medical interventions, influenza can be associated with pneumonia and even death, especially in the very young, the elderly, and persons with underlying medical conditions such as pulmonary, cardiovascular, renal, and liver diseases [Paules 2017].

Influenza viruses are enveloped viruses belonging to the family of Orthomyxoviridae and are divided into 3 types, designated A, B, and C. Type A and B influenza viruses are responsible for yearly epidemic outbreaks of respiratory illness. Type A influenza viruses are further subdivided into subtypes based on the antigen structure of the 2 major surface glycoproteins, hemagglutinin (HA) and neuraminidase (NA). Among influenza A viruses, 18 HA subtypes and 11 NA subtypes are known to exist in viruses circulating among wild waterfowl. However, at this time, viruses characterized by only 2 combinations of HA and NA subtypes, H1N1 and H3N2, are stably established and circulate widely among humans, although H2N2 and H3N8 viruses have been established in humans in the past [Paules 2017]. Unlike Type A, Type B viruses are restricted to humans. Currently, 2 influenza B virus genetic lineages are in co-circulation. These lineages, termed Yamagata and Victoria based on their prototype strains, have limited antigenic cross-reactivity and often circulate together during the yearly epidemic [Paules 2017].

# 1.2 Influenza Disease Burden in Older Adults

Older adults are at the greatest risk of hospitalization and death due to influenza infection [CDC 2019b]. A retrospective study of 3 managed-care organizations during 1996 to 1997 through 1999 to 2000 estimated that the incidence rate of hospitalization during influenza season among people ≥ 65 years of age with underlying high-risk conditions was 55.6 pneumonia and influenza-associated hospitalizations per 10,000 persons, compared with 18.7 per 10,000 among lower-risk people of the same age group. Older adults between the ages of 50 to 64 with underlying conditions were also at increased risk for hospitalization during influenza seasons (12.3 per 10,000), compared with healthy older adults (1.8 per 10,000) [Mullooly 2007]. Between the years 1976 to 2007, approximately 21,098 older adults (≥ 65 years) were estimated to have died annually due to an influenza-related cause, corresponding to 90% of estimated annual average influenza-related mortality across all age groups [CDC 2010]. Data from modeling analyses of population-based surveillance covering 2010 to 2011 through 2012 to 2013 influenza seasons suggests that 71 to 85% of all influenza-related deaths occurred in adults > 65 years of age [Reed 2015, Grohskopf 2016].

# 1.3 Licensed Vaccines Against Influenza Virus for Older Adults

Vaccination is the cornerstone of influenza control, particularly for high-risk individuals older than 65 years, immunocompromised patients, and young children; and offers the most cost-effective approach to reduce the morbidity, mortality, and economic burden associated with influenza infection [Paules 2017]. To date, 7 quadrivalent inactivated or recombinant influenza vaccines, consisting of 2 A virus strains (A/H3N2 and A/H1N1) and strains of both B lineages, are licensed for sale in the US and marketed for the 2018-19 influenza season, indicated for various populations [FDA 2019, CDC 2019a]. These include the egg-derived inactivated virus vaccines Afluria® (Seqirus), Fluarix® (GlaxoSmithKline), FluLaval® (ID Biomedical Corp. of Quebec), Fluzone® (Sanofi Pasteur), and Fluzone intradermal (Sanofi Pasteur); the cell culture-derived vaccine Flucelvax® (Seqirus), and the recombinant DNA technology-derived Flublok® Quadrivalent (Sanofi Pasteur, previously Protein Sciences). Three trivalent inactivated or recombinant influenza vaccines are also approved and marketed for the 2018-19 influenza season in the US [CDC 2019a]. Only 1 influenza vaccine is approved with an adjuvant (FLUAD<sup>TM</sup> with adjuvant MF59) [CDC 2019a].

Of all currently-licensed vaccines, 2 are specifically approved for use in older adults, and include a high-dose (ie, Fluzone® High-Dose [Fluzone HD] initially approved in the US in 2009) and an adjuvanted standard-dose inactivated vaccine (ie, FLUAD initially approved in the US in 2015); both of these are trivalent [CDC 2019a]. There are currently no data available that compare the immunogenicity of FLUAD to Fluzone HD in a randomized clinical trial. Although Fluzone HD has reported an increased relative vaccine efficacy of approximately 24% in the older adult population compared with standard-dose Fluzone [DiazGranados 2014, Monto 2017], effectiveness rates reported in older adults have remained quite variable, though uniformly suboptimal, from season-to-season since the approval of Fluzone HD in 2009, ranging anywhere from -5.8% to 45% from 2009 to 2018 [Griffin 2011, Treanor 2012, Ohmit 2014, Reed 2014, McLean 2015, Flannery 2018, Zimmerman 2016, CDC 2019a]. During the current influenza season (2018 - 19), interim estimates indicate that vaccine efficacy in older adults (≥ 50 years of age) remains relatively low at 24% (-15% to 51%) against all influenza types [Doyle 2019]. This variability is multifactorial, but is likely, in part, due to antigenic drift or mismatch between circulating and vaccine influenza strains leading to reduced effectiveness of seasonal influenza vaccines. The most recent example of unanticipated drift occurred in the Northern hemisphere 2014-15 influenza season, when A(H3N2) clade 3C.2a viruses replaced A/Texas/50/12-like clade 3C.1 viruses represented in the vaccines. This mismatch between vaccine and circulating viruses resulted in vaccine effectiveness not different from zero [Skowronski 2016]. Emerging data also demonstrate other mechanisms that may account for reduction in vaccine effectiveness, specifically the increasingly-recognized problem of antigenic changes arising from egg-based influenza vaccine production. It has been shown that hemagglutinin proteins produced by viruses replicating in eggs undergo adaptive mutations which can critically alter the antigenic structure of key HA head-based epitopes and consequently, the immune response in the vaccinee and thereby result in an apparent antigenic mismatch between egg-produced vaccine strains and circulating strains [Zost 2017]. This mechanism, compounded by a degree of antigenic evolution, may explain the very poor effectiveness of 2017 vaccines against A(H3N2) viruses in Australia [Sullivan 2017]. Thus, there remains a significant need for influenza vaccines with improved efficacy, and, in

particular, the capacity to mitigate the consequences of both naturally-occurring antigenic drift between strain selection and circulation of the virus, as well as, potential egg-adaptive mutations giving rise to deleterious antigenic changes. The need for improved vaccine performance is the greatest in the older adult population, which remains vulnerable to serious complications, including death, resulting from influenza infection. Accordingly, a vaccine which induces both strong homologous, as well as broadly cross-reactive, hemagglutination inhibition (HAI) antibodies, induces potent broadly cross-reactive strain-specific polyfunctional CD4+ T cell responses, and is produced in a recombinant wild-type expression system (thereby avoiding the problem of egg adaptive mutations), could be of significant added value and could help meet the unmet medical need of influenza prevention in older adults.

# 1.4 Novavax's Nanoparticle Influenza Vaccines

# 1.4.1 Quadrivalent (Quad-NIV)

Novavax's Quad-NIV is based on purified, recombinant, full-length HA that self-assemble into distinct nanoparticle structures of approximately 20 to 40 nm [Smith 2017]. A baculovirus/Spodoptera frugiperda (Sf9) insect cell system is used to clone and express recombinant influenza HAs from the 4 influenza strains recommended for the relevant influenza season. For the 2019 - 20 Northern Hemisphere influenza season, strains include: A/Brisbane/02/2018 (H1N1) pdm09; A/Kansas/14/2017 (H3N2); B/Maryland/15/2016 (Victoria lineage); and B/Phuket/3073/2013 (Yamagata lineage) [VRBPAC 2019, WHO 2019].

# 1.4.2 Trivalent (Tri-NIV)

Novavax had previously also developed Tri-NIV, a trivalent precursor to Quad-NIV, which was based on purified, recombinant, full-length HA that self-assembles into distinct nanoparticle structures of approximately 20 to 40 nm [Smith 2017], and manufactured using the same Sf9 technology used to manufacture Quad-NIV. Tri-NIV comprised recombinant influenza HAs from influenza strains recommended for the 2017-18 Northern Hemisphere influenza season: A/Michigan/45/2015 (H1N1); A/HongKong/4801/2014 (H3N2); and B/Brisbane/60/2008 [WHO 2017].

Summaries of non-clinical and clinical data for Tri-NIV are available in Section 1.5.1 and in the Investigator's Brochure (IB), respectively.

# 1.4.3 Matrix-M1 Adjuvant

Adjuvants are compounds which, when combined with a specific vaccine antigen, serve to increase the immune response to the vaccine. In general, adjuvants work by engaging one or more components of the innate immune system, a system that provides a rapid response to infection or tissue damage based on recognition of molecular structures common to large groups of microbial pathogens [Coffman 2010]. Thus, adjuvants may both quantitatively increase the antibody response and also qualitatively broaden its specificity. In addition, some adjuvants may modulate the cellular immune response.

Matrix-M1 is a saponin-based adjuvant, which can be co-administered with an antigen to induce a targeted immune response. Matrix-M1 is manufactured by mixing defined, partially-purified

extracts of the bark of the *Quillaja saponaria* Molina tree with cholesterol and phosphatidylcholine in the presence of a detergent. Removal of detergent by diafiltration results in the formation of stable cage-like structures of 2 types, designated Matrix-A and Matrix-C, dependent on the precise *Quillaja* extract incorporated. Matrix-A and -C are blended in an 85:15 ratio, respectively, to yield Matrix-M1. The proposed mode of action of Matrix-M1 does not include a depot effect, but rather is through a combination of activities including recruitment and activation of innate immune cells, rapid antigen delivery to antigen presenting cells (APCs), and enhanced antigen presentation via both Major Histocompatibility Complex (MHC) I and MHC II molecules in the draining lymph nodes.

# 1.5 Nonclinical Investigations

# 1.5.1 Matrix-M1-adjuvanted Tri-NIV

A key animal study of Tri-NIV, a trivalent precursor to Quad-NIV (see Section 1.4.2), was conducted in an influenza disease model (ferrets) to evaluate its immunogenicity and protective efficacy against both a recent and drifted A/H3N2 challenge strain; and to compare the immune response with that of the 2016-17 Fluzone HD and Fluzone Quadrivalent (standard dose) vaccines. In ferrets, Tri-NIV administered with Matrix-M1 adjuvant elicited rapid and robust immune responses in terms of geometric mean hemagglutinin inhibition (HAI) titers, with responses exceeding those induced by Fluzone HD or Fluzone Quadrivalent. Secondly, geometric mean 50% microneutralizing (MN) titers against a broad panel of historic H3N2 strains tested, dating to 1999 and spanning a number of clinically-significant antigenic drift events, showed 2 to 214-fold higher titers among animals given Tri-NIV with Matrix-M1 adjuvant than among animals given Fluzone HD. These data suggest that Tri-NIV may elicit antibodies to broadly-neutralizing epitopes capable of providing greater antigenic drift strain protection, even against strains such as A/HongKong/4801/2014, which are associated with impaired influenza vaccine efficacy in humans.

Additionally, a good laboratory practices (GLP)-compliant, repeat-dose toxicology study was conducted in New Zealand White (NZW) rabbits investigating the safety and immunogenicity of a total dose of 60 µg of a nanoparticle influenza vaccine (NIV), a precursor to Tri-NIV (containing 30 µg each of A/Switzerland/9715293/2013 and B/Brisbane/60/2008 [in addition to A/Anhui/1/2013 neuraminidase alone or in combination with RSV F protein, which are not present in the current candidate], and generated using the same baculovirus/Sf9 technology as Tri-NIV and Quad-NIV) was administered to animals on Days 1 and 15, alone or with 50 µg Matrix-M1 adjuvant. Results showed no adverse effects on mortality, physical examinations, cageside observations, dermal Draize observations, body weights, body weight changes, food consumption, body temperatures, ophthalmology, clinical chemistry, hematology, gross pathology, or histopathology, with robust influenza-specific responses observed among actively-immunized animals, when compared to placebo. There were mild inflammatory responses at the vaccine injection sites and hyperplasia of the lymph nodes draining the injection sites, which were accompanied by elevation of serum inflammatory markers (eg, CRP and fibrinogen). These effects were transient and showed rapid resolution and were considered normal, non-adverse responses to immunization. A complete description of these nonclinical studies is provided in the IB.

### 1.5.2 Other Matrix-M1-adjuvanted Vaccines

Additional toxicological studies in NZW rabbits have been performed with two different antigens, ie, an influenza virus (H7N9) virus-like particle and an Ebola virus glycoprotein, in which up to 100 µg Matrix-M1 alone or with antigen was evaluated. These toxicological investigations indicated that Matrix-M1 adjuvant in doses up 100 µg was well-tolerated in the animal and antigen system tested with no evidence of toxicity suggestive of any unusual risk or target organ for toxicity. Non-adverse findings, including local injection site reactions and chemical markers of inflammation, were transient and similar to those reported in the NIV toxicology study and were considered consistent with immune system stimulation consequent to immunization. Reference the Matrix-M<sup>TM</sup> Adjuvant Safety Data Supplement for details regarding these additional toxicology studies.

# 1.6 Clinical Investigations

# 1.6.1 Summary of Phase 2 Trial (qNIV-E-201) with Quad-NIV

In a Phase 2, randomized, observer-blinded, active-controlled trial (qNIV-E-201), Novavax evaluated the safety and immunogenicity of various formulations (antigen doses) of Quad-NIV, based on the four 2018 - 19 Northern Hemisphere influenza season strains: A/Michigan/45/2015 (H1N1); A/Singapore/INFIMH-16-0019/2016 (H3N2); B/Colorado/06/2017; and B/Phuket/3073/2013, in adults  $\geq$  65 years of age (n = 1375 subjects), administered alone or with Matrix-M1 adjuvant compared with Fluzone® High-Dose (HD) and Flublok® Quadrivalent. Safety and immunogenicity results through Day 28 are available and briefly summarized below.

# 1.6.1.1 Safety Through Day 28

Overall, various formulations (antigen/adjuvant doses) of Quad-NIV administered alone or with Matrix-M1 adjuvant showed an acceptable safety profile and were well-tolerated, with no significant dose-related toxicities observed. The proportion of subjects with AEs was comparable across all adjuvanted Quad-NIV groups (41 - 52%) and the active comparators, Fluzone HD (47%) and Flublok (44%); AEs were reported slightly less frequently in the unadjuvanted Quad-NIV group (38%). It is notable that the safety profile of Quad-NIV remained comparable across groups regardless of increasing the total antigen dose (ie, total HA of 180  $\mu$ g in Phase 1/2 vs 240 or 300  $\mu$ g HA in Phase 2) or adjuvant dose (ie, 50 or 75  $\mu$ g Matrix-M1). Further, the safety profile of Quad-NIV formulated with the Matrix-M1 adjuvant remained comparable to the unadjuvanted active comparators used in this trial.

Note: The following individual safety summaries regarding solicited and unsolicited AEs, MAEs, and SAEs pertain to subjects who received 240  $\mu$ g of Quad-NIV co-formulated with 75  $\mu$ g Matrix-M1, as compared to those who received Fluzone HD or Flublok, as this is the dose and formulation selected for evaluation in the present Phase 3 trial.

Solicited AEs (common vaccine reactogenicity complaints occurring in the first 7 days after exposure) occurred with similar frequency in the 240 µg Quad-NIV with 75 µg Matrix-M1 group (38%) compared with the Fluzone HD and Flublok groups (37 - 38%). These events included typical transient vaccine reactogenicity complaints, and all were transient. It is noted

that a slightly higher frequency of severe solicited AEs occurred among Quad-NIV recipients (3.2%) as compared with Fluzone HD recipients (1.3%) and to a lesser extent Flublok (2.6%); however, the 95% confidence intervals were overlapping among all groups. Severe fever was not reported in any treatment group.

Unsolicited AEs were reported by similar proportions of subjects who received 240  $\mu g$  Quad-NIV with 75  $\mu g$  Matrix-M1 (18%) and Fluzone HD (20%), and slightly less in the Flublok group (15%), through Day 28. Reports of severe unsolicited AEs were uncommon and reported in 2% of subjects in the Quad-NIV group and 1% of subjects in each of the active comparator groups. One severe event each of blood urea increased, anxiety, and nephrolithiasis was reported in the Quad-NIV group (3/156 subjects); acute sinusitis, dehydration, and hypokalemia in the Fluzone HD group (1/153 subjects); and hypertension in the Flublok group (1/151 subjects); none of these events were reported by the investigator as related to study treatment.

MAEs were reported in a similar proportion of subjects across all groups (7% Quad-NIV [240 µg HA with 75 µg Matrix-M1]; 9% Fluzone HD; 6% Flublok) with diagnoses spanning several SOCs, most commonly infections and infestations, representing common intercurrent illnesses with no apparent clustering by treatment group. SNMCs were reported in 2% of Quad-NIV subjects and 1% of Fluzone HD and Flublok subjects. Similar to MAEs, the diagnoses span several SOCs representing common intercurrent illnesses in this older adult population with no apparent clustering by treatment group.

No serious adverse events (SAEs) leading to death or considered related to study treatment have been reported to date. SAEs were reported in one subject each in the 240  $\mu g$  Quad-NIV with 75  $\mu g$  Matrix-M1 group (malignant melanoma) and the Fluzone HD (dehydration) group; no SAEs have been reported to date in the Flublok group. Generally, the rate of SAEs is consistent with the rate of 1.3% within 30 days post-vaccination reported in the Fluzone HD USPI (June 2018).

Overall, the safety and reactogenicity profiles of various formulations of Quad-NIV were generally comparable to both active comparator influenza vaccines based on available data through Day 28.

### 1.6.1.2 Immunogenicity Through Day 28

Overall, immunogenicity results demonstrated that all Matrix-M1 adjuvanted formulations of Quad-NIV were immunogenic, inducing robust HAI responses against homologous A and B influenza strains, as well as against drifted A/H3N2 strains (A/Switzerland/9715293/2013 and A/Wisconsin/19/2017). Moreover, all Matrix-M1 adjuvanted formulations of Quad-NIV were generally at least comparable to both Fluzone HD and Flublok using the egg-propagated virus or wild-type virus-like particle (VLP) HAI assay formats. Importantly, all Matrix-M1 adjuvanted formulations of Quad-NIV had significantly greater HAI responses compared with Fluzone HD for A/H3N2 strains, both homologous and drifted, as evaluated in the wild-type VLP-based HAI assay. These Quad-NIV formulations were comparable or better than Fluzone HD (not statistically significant) against these same A/H3N2 strains in the egg-propagated assay. Several formulations of Matrix-M1 adjuvanted Quad-NIV were significantly lower for

B/Colorado/06/2017 in the egg-propagated HAI assay compared with Fluzone HD, but remained comparable (ie, no significant difference) in the VLP-based assay. However, it should included noted that both Fluzone HD and Flublok B/Maryland/15/2016 (a B/Colorado/06/2017-like virus) for the Victoria lineage B strain in their 2018 - 19 vaccine formulations used in this trial, rather than the B/Colorado/06/2017 strain used in the Quad-NIV formulations. While both strains were recommended by WHO as acceptable alternative "like" strains for the B Victoria lineage, the B/Maryland/15/2016 strain systematically induced 2-fold higher HAI antibody responses compared to B/Colorado/06/2017 in ferret studies reported by the CDC and WHO [VRBPAC 2018].

In terms of cell-mediated immunity (CMI), several Matrix-M1 adjuvanted formulations of Quad-NIV induced potent strain-specific and cross-reactive polyfunctional CD4+ T cell responses. Lastly, as described in further detail in Section 1.7, these safety and immunogenicity data support further clinical development of Quad-NIV with Matrix-M1 adjuvant (60 µg per HA strain co-formulated with 75 µg of Matrix-M1 adjuvant) in this Phase 3 clinical trial given that increasing the Matrix-M1 adjuvant dose from 50 µg to 75 µg appeared to further enhance polyfunctional CD4+ T cell responses while maintaining comparable HAI responses and a comparable safety profile relative to formulations of Quad-NIV containing 50 µg of Matrix-M1.

### 1.6.2 Matrix-M-adjuvanted Vaccines

Matrix-M adjuvant, in 1 of 2 formulations (ie, Matrix-M1 and Matrix-M2), has been administered with a variety of vaccine antigens to over 2350 human subjects in multiple clinical trials in the US, Europe, and Australia. Of this, over 1800 subjects have received vaccines containing the Matrix-M1 adjuvant (proposed for use in this trial) and 537 subjects have received vaccines containing Matrix-M2 adjuvant (an adjuvant containing the same active components as Matrix-M1, but in a slightly different ratio). Among all 15 studies, no reported serious adverse events (SAE) have been classified as related to exposure to the Matrix-M adjuvant.

Please refer to the most recent version of the Matrix-M<sup>TM</sup> Adjuvant Safety Data Supplement for detailed summaries of the clinical experience with Matrix-M1-adjuvanted vaccines.

#### 1.7 Trial Rationale

The influenza virus poses a formidable risk of infection resulting in serious illness in older adults. Based on estimates by the Centers for Disease Control and Prevention (CDC), in the US alone, up to 85% of all influenza-related deaths and 70% of all influenza-related hospitalizations occur in people 65 years of age or older [CDC 2017]. During the current influenza season (2018 - 19), interim estimates indicate that vaccine efficacy in older adults ( $\geq$  50 years of age) remains relatively low at 24% (-15% to 51%) against all influenza types [Doyle 2019]. In light of the continued suboptimal effectiveness of seasonal influenza vaccines, particularly in older adults.

Novavax has developed a novel recombinant hemagglutinin (HA) quadrivalent nanoparticle influenza vaccine (Quad-NIV) for the prevention of disease due to influenza virus in adults  $\geq 65$  years of age, using a recombinant baculovirus and insect cell technology. With a

nanoparticle structure, recombinant wild-type sequenced HAs, and use of Matrix-M1 adjuvant, Quad-NIV may offer several important advantages over existing licensed egg-derived seasonal influenza vaccines, including avoidance of antigenic mismatch due to egg-adaptive mutations; induction of both broadly cross-reactive antibody responses against emerging drift variants of seasonal influenza viruses [Shinde 2018]; and potent cross-reactive polyfunctional CD4+ T cells.


In a recent Phase 2, dose-finding, formulation-optimizing trial in adults  $\geq 65$  years of age, multiple formulations of Quad-NIV, containing HA-based antigens representing the 4 influenza strains recommended for inclusion in the 2018 - 2019 Northern hemisphere seasonal influenza vaccine [VRBPAC 2018, WHO 2018] and co-formulated with Matrix-M1 adjuvant, given intramuscularly, induced robust hemagglutination inhibition (HAI) antibody responses against both homologous A/B and drifted H3N2 strains. Three formulations in particular: formulation A (60 μg HA of each strain in-clinic mixed with 50 μg of Matrix-M1); formulation B (60 μg HA of each strain co-formulated with 50 µg of Matrix-M1); and formulation C (60 µg HA of each strain co-formulated with 75 µg of Matrix-M1), induced comparable HAI antibody responses (using both egg-propagated or wild-type VLP agglutinins as reagents) against all evaluated homologous and drifted H3N2 strains. In addition, all three formulations outperformed Fluzone HD on HAI antibody responses to all evaluated homologous and drifted H3N2 strains using the wild-type VLP HAI assays, which assessed the binding of vaccine-induced antibodies to HA sequences reflective of circulating viruses not subjected to egg adaptation. The short-term reactogenicity and overall safety profiles (through 182 days of follow-up) of the three formulations were also comparable. Formulation C (60 µg HA of each strain co-formulated with 75 µg of Matrix-M1) induced substantially higher median counts of homologous and drifted strain-specific polyfunctional CD4+ T cells at Day 7 following immunization. Finally, formulation C elicited significantly higher mean hemagglutination inhibition (HAI) titers than unadjuvanted Quad-NIV (formulation E containing only 60 µg HA of each strain) for 5 of 6 tested viral hemagglutinins. The totality of safety and immunogenicity data to date indicate that formulation C of Quad-NIV is the best candidate to advance in further clinical development.

The Phase 2 data warrant confirmation of the non-inferiority of immunogenicity of 240 µg Quad-NIV containing antigens (60 µg HA of each strain) representing the 4 influenza strains recommended for inclusion in the 2019 - 2020 Northern hemisphere seasonal influenza vaccine [VRBPAC 2019, WHO 2019], co formulated with 75 µg Matrix-M1 adjuvant, as compared to a US-licensed quadrivalent seasonal influenza vaccine comparator, Fluzone Quadrivalent, to generate data to support licensure of Quad-NIV for the prevention of influenza disease in adults  $\geq$  65 years of age.

#### **Expected Risks from Vaccination with Quad-NIV With or Without** 1.8 Matrix-M1 Adjuvant

The expected risk of vaccination with Quad-NIV in combination with Matrix-M1 adjuvant can be directly extrapolated from available safety data through Day 28 from the previous Phase 2 trial (qNIV-E-201), which tested Quad-NIV alone or adjuvanted with Matrix-M1 in adults  $\geq$  65 years of age (n = 1375 subjects) compared with Fluzone HD and Flublok Quadrivalent. To date, there have been a total of 1068 human exposures to Quad-NIV with or without Matrix-M1 adjuvant.

Overall, the safety and reactogenicity profile of all Quad-NIV formulations/groups have been generally comparable to the active comparator influenza vaccines (Fluzone HD and Flublok Quadrivalent) based on available data reviewed through Day 28. A slightly higher frequency of severe solicited AEs occurred among subjects who received 240 µg Quad-NIV with 50 µg Matrix-M1 (3.3%) or 240 µg Quad-NIV with 75 µg Matrix-M1 (3.2%) relative to the active comparators (delta of < 1%); however, the 95% confidence intervals were overlapping among all groups. Injection site pain was the most common local AE (19%) followed by swelling (7%). In the group that received 240 µg Quad-NIV with 75 µg Matrix-M1, the most common systemic AEs (> 10%) were headache (15%) and muscle pain (10%). Reports of respiratory/facial AEs were generally infrequent and occurred in  $\leq 5\%$  of subjects, with the exception of cough and sore throat, which occurred in 8% of subjects. Severe events occurring in subjects who received 240 µg Quad-NIV with 75 µg Matrix-M1 included nausea, fatigue, headache, sore throat, diarrhea, vomiting, chills, joint pain, muscle pain, difficulty swallowing, and eye redness, although these did not occur in significantly greater proportions than in subjects who received Fluzone HD or Flublok. Persistence of these signs and symptoms beyond 7 days after injection occurs uncommonly and is not expected. Occurrence of these solicited signs and symptoms with characteristics consistent with the definition of a SAE (ie, need for an urgent and significant medical intervention, and/or hospitalization, and/or residual disability) is also not expected.

Finally, risks identified in human clinical trials with the Matrix-M1 adjuvant have been described in detail in the current Matrix-M Adjuvant Safety Data Supplement, which is provided for information with the protocol and the Quad-NIV Investigator's Brochure.

#### 1.9 Risks Associated with Fluzone Quadrivalent

In adults  $\geq$  65 years of age, the most common ( $\geq$  10%) injection-site reaction was pain (33%) and the most common solicited systemic adverse reactions were myalgia (18%), headache (13%), and malaise (11%). Unsolicited non-serious adverse events were reported in 12.4% of recipients in the Fluzone Quadrivalent group, as compared to 9.8% of recipients in either of the comparator trivalent influenza vaccine groups (TIV-1 or TIV-2). The most commonly reported adverse events were oropharyngeal pain, rhinorrhea, injection-site induration, and headache.

Information regarding the post-marketing safety data for Fluzone Quadrivalent is available in the Package Insert, which will be supplied to Investigators. Of note, subjects with a history of Guillain-Barré syndrome within 6 weeks of any influenza vaccine should not receive Fluzone Quadrivalent or be enrolled in this trial (see trial exclusion criteria in Section 5.2).

# 2 TRIAL OBJECTIVES

# 2.1 Primary Objectives

- To demonstrate the non-inferior immunogenicity of 240 μg Quad-NIV co-formulated with 75 μg Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of hemagglutination inhibition (HAI) (assayed with egg-propagated virus) antibody responses to all Quad-NIV homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) at Day 28 post-vaccination.
- To describe the safety profile of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, and the comparator in clinically stable adults ≥ 65 years of age. The safety profile will include solicited short-term reactogenicity; 28-day all adverse event (AE) profile; 1-year post-injection medically-attended adverse event (MAE), serious adverse event (SAE), and significant new medical condition (SNMC), including immunologically-mediated adverse events of special interest (AESIs).

# 2.2 Secondary Objectives

• To describe the immunogenicity of 240 μg Quad-NIV co-formulated with 75 μg Matrix-M1 adjuvant, and of a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of HAI (assayed with both egg-propagated virus and wild-type VLP reagents) antibody responses to all Quad-NIV homologous influenza strains (2 influenza A and 2 influenza B strains) and at least 1 antigenically drifted A or B strain in terms of geometric mean titers (GMTs), geometric mean ratio (GMR), seroconversion rate (SCR), seroprotection rate (SPR), and the baseline adjusted ratio of GMTs between treatment arms at Day 28. An additional time-point at Day 182 may be tested by HAI for these outcomes in a subset of subjects in each treatment group.

# 2.3 Exploratory Objectives

- To evaluate the superior immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, relative to Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of HAI (assayed with both egg-propagated virus and wild-type VLP reagents) antibody responses against all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and 1-2 antigenically-drifted A and/or B strains at Days 0 and 28 post-vaccination.
- To describe the immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, and of a US-licensed comparator, Fluzone Quadrivalent, in clinically stable adults ≥ 65 years of age, in terms of microneutralization (MN) responses to vaccine-homologous and/or antigenically-drifted influenza strains at Days 0 and 28 post-vaccination, in terms of GMTs, GMR, SCR, and the baseline adjusted ratio of GMTs between treatment arms at Days 28 post-vaccination. *Note: Due to the time-consuming nature of MN testing, this exploratory objective may be completed in a subset of participants in each study treatment group and/or a subset of strains after the initial study HAI data are complete and reported in an addendum. Laboratory staff will remain blinded as to treatment assignments until all projected MN tests are complete. Similarly, an additional time-point at Day 182 may also be tested.*

• To describe the quality and amplitude of cell-mediated immune (CMI) responses in healthy adults  $\geq$  65 years of age to vaccination with 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, as measured by functional T cell responses based on intracellular cytokine analysis. Additional markers of CMI (eg, memory B cells and/or other T cell subsets) may be evaluated depending on availability/recovery of cell volume. Due to the laborious nature of the cellular assays, they will be performed on subjects from a limited number of participating sites and results may be reported as an addendum to the main clinical study report.

#### 3 TRIAL OVERVIEW

# 3.1 Design

This is a Phase 3, randomized, observer-blinded, active-controlled trial to evaluate the immunogenicity and safety of 240  $\mu$ g Quad-NIV co-formulated with 75  $\mu$ g Matrix-M1 adjuvant against a licensed comparator in clinically stable adults  $\geq$  65 years of age to be conducted in the United States. Approximately 2650 eligible subjects will be enrolled and randomized at a 1:1 ratio into 1 of 2 treatment groups, as shown in Table 1 below. The active group (Group A) and the comparator group (Group B) will each consist of approximately 1325 subjects. Both groups will be stratified by site, age (65 to < 75 and  $\geq$  75 years), and history of prior year receipt of the 2018 - 19 influenza vaccine. On Day 0, all subjects will receive a study treatment as indicated in Table 1 by intramuscular (IM) injection. Total injection volumes for Quad-NIV will be 0.5 mL. Trial follow-up for each subject will span approximately 1 year from the Day 0 injection. It is anticipated that a percentage of the randomized trial subjects will not complete the trial. Subjects who withdraw or are discontinued will not be replaced.

Table 1: Trial Design for qNIV-E-301

| | | Day 0 Trial Treatme | | | | |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Vaccine HA Dose per Strain, μg (H1N1/H3N2/B <sub>V</sub> /B <sub>Y</sub> ) Matrix-M1 Adjuvant Dose Volume | | | | Treatment<br>Arm | Subjects Per<br>Group |
| A | Quad-NIV | 60, 60, 60, 60 | 75 µg | 0.5 mL | Non-dominant | 1325 |
| В | | 2019-20 Fluzone Qu | ıadrivalent <sup>[1]</sup> | | Non-dominant | 1325 |
| Total Trial Subjects | | | | | 2650 | |

Abbreviations:  $B_V = B$  Victoria lineage;  $B_Y = B$  Yamagata lineage; HA = Hemagglutinin

Note: All subjects will receive a single vaccination by IM injection on Day 0. If the non-dominant arm is not available for injection, then the dominant arm will be used.

# 3.2 Trial Endpoints

# 3.2.1 Primary Endpoints

- Comparative HAI antibody responses (assayed with egg-propagated virus) on Day 28, summarized in terms of the ratio of geometric mean titers (GMTs) AND seroconversion rate (SCR) difference, between subjects receiving Quad-NIV or Fluzone Quadrivalent for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains). Non-inferiority for each homologous strain will be demonstrated if:
  - $\circ$  The lower bound of the two-sided 95% CI on the ratio of the GMTs (GMT\_{QuadNIV}/GMT\_{Fluzone}) is  $\geq 0.67,$

### AND

○ The lower bound of the two-sided 95% CI on the difference between the SCRs ( $SCR_{QuadNIV}$ - $SCR_{Fluzone}$ ) is  $\geq$  -10%.

<sup>[1]</sup> Fluzone Quadrivalent will be administered at the manufacturer's recommended dose and volume.

• Number and percentage (95% CI) of subjects with solicited local and systemic adverse events over the 7 days post-injection (ie, Day 0 through Day 6, inclusive); all adverse events through 28 days post-injection (ie, Day 0 through Day 27, inclusive); and MAEs, SAEs, and SNMCs – including AESIs – through 1 year post-injection.

# 3.2.2 Secondary Endpoints

- HAI antibody titers (assayed with both egg-propagated virus and wild-type VLP reagents) at Days 0 and 28 specific for vaccine-homologous A and B strain(s), and antigenically-drifted influenza strains. An additional time-point at Day 182 may also be tested with a subset of subjects. Derived/calculated endpoints based on these data will include:
  - o GMT defined as the antilog of the mean of the log-transformed HAI titers, on Days 0 and 28.
  - o Geometric mean ratio (GMR) defined as the ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs (GMR<sub>Post/Pre</sub>) on Day 28.
  - O Seroconversion rate (SCR) defined as proportion of subjects in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer  $\ge 40$ , or a baseline reciprocal (Day 0) titer of  $\ge 10$  and a post-vaccination titer  $\ge 4$ -fold higher on Day 28.
  - $\circ$  Seroprotection rate (SPR) defined as the proportion of subjects with a reciprocal HAI titer  $\geq$  40 on Day 28.
  - o Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).

# 3.2.3 Exploratory Endpoints

Comparative HAI antibody responses (assayed with both egg-propagated virus and wild-type VLP reagents) on Day 28, summarized in terms of the ratio of geometric mean titers (GMTs) AND seroconversion rate (SCR) difference, between subjects receiving Quad-NIV or Fluzone Quadrivalent for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and 1 - 2 antigenically-drifted A and/or B strains.

Superior immunogenicity for each strain will be demonstrated if:

 $\circ$  The lower bound of the two-sided 95% CI on the ratio of the GMTs (GMT<sub>OuadNIV</sub>/GMT<sub>Fluzone</sub>) is greater than 1.5,

#### AND

- The lower bound of the two-sided 95% CI on the difference between the seroconversion rates (SCR<sub>QuadNIV</sub>-SCR<sub>Fluzone</sub>) is greater than 10%.
- Microneutralization (MN) responses: Neutralizing antibody titers specific to vaccine-homologous A and B strain(s) and/or antigenically-drifted influenza strains, at Days 0 and 28 post-vaccination, as measured by a microneutralization assay. An additional time-point at Day 182 may also be tested. Derived/calculated endpoints based on these data will include:

- GMT defined as the antilog of the mean of the log-transformed neutralizing titer for a given treatment group.
- o GMR defined as the ratio of post-vaccination and pre-vaccination neutralizing GMTs within the same treatment group (designated as GMR<sub>Post/Pre</sub>).
- o SCR defined as proportion of subjects in a given treatment group with either a baseline reciprocal titer of < lower limit of quantitation (LLOQ) and a post-vaccination reciprocal titer 4-fold higher than the LLOQ, or a baseline reciprocal titer of ≥ LLOQ and a post-vaccination reciprocal titer ≥ 4-fold higher than the baseline titer.
- o Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).
- Counts and/or proportions of Days 0, 7, 28, and 182 peripheral blood effector memory T cell populations that secrete one or more of IL-2, CD40L, IFN-γ, and TNF-α cytokines following *in vitro* restimulation with HA in subjects selected for cellular immune response monitoring. Counts and/or proportions of additional markers of CMI, as appropriate.

# 3.3 Randomization and Blinding Procedure

Subject randomization will be conducted using an Interactive Web Randomization System (IWRS). Stratification will be by site, age, and history of receipt of the 2018-19 influenza vaccine. Proportions of subjects in the various strata will not be pre-specified; rather, the goal will be to achieve an approximately equal distribution of subjects with these characteristics across the two treatment groups.

Preparation and administration of each test article dose will be performed by unblinded vaccine pharmacists/administrators. These persons, identified prior to trial dosing, will not perform any trial assessments post-dosing.

# 3.4 Maintaining the Blinded Randomization Scheme

Randomization procedures will be performed using IWRS, with treatment assignments known only to the responsible unblinded vaccine administrators at the trial center. Subjects and the main trial team clinical staff will remain blinded for the duration of the trial unless emergency unblinding is necessary. Refer to Section 3.5 for information regarding the process for emergency unblinding.

All treatment assignments, vaccine storage and accountability, and/or dosing-related matters will be monitored by a designated "unblinded monitor." Any deviations will be discussed, documented, and resolved by the unblinded monitor and the unblinded site personnel. Reports provided by the unblinded monitor will be reviewed by designated unblinded personnel at either Novavax or the clinical research organization (CRO), not involved with the main trial team. No reports from the unblinded monitor will be released to the Trial Master File (TMF) until database lock for Day 364.

# 3.5 Procedure for Unblinding Individual Subjects During the Trial

In the event of a medical emergency, when knowledge of one or more subject's treatment assignment may influence his/her clinical care or the conduct of the trial, the sponsor's Chief

Medical Officer (CMO) or an investigator or designee may request that the blind be broken for the subject(s) experiencing the emergency. Prior to unblinding for individual subjects at site investigator's request, however, the requesting party must use all reasonable efforts to contact the Medical Monitor or designee to discuss the decision to break the blind. In the case of such individual subjects, the investigator will be expected to provide a rationale for the necessity of unblinding based on a meaningful change to the subject's immediate and short-term medical care which will result from knowledge of treatment assignment.

Novavax retains the right to unblind the treatment allocation for SAEs that are unexpected and are suspected to be causally related to the test article, and that potentially require expedited reporting to regulatory authorities.

If unblinding of an individual subject is deemed necessary, the unblinded staff member shall obtain subject dose details from the randomization system. The date and time of breaking the blind as well as the reason must be recorded and placed in the Pharmacy Binder by unblinded staff. The individual subject dose details should be revealed only in case of an emergency where further treatment of the subject is dependent on knowing the investigational product he/she has received. The investigator should not otherwise divulge the subject's treatment assignment to site staff, and should provide the information only to those individuals involved in the direct care of the subject. The date and reasons for breaking the blind must be submitted to the Medical Monitor within 24 hours.

### 3.6 Trial Duration

The maximum duration of an individual subject's participation in the trial conduct is approximately 1 year.

#### 4 TRIAL TEST ARTICLES

The investigational product (IP) under evaluation in this trial is Quad-NIV adjuvanted with Matrix-M1 adjuvant. Discussions on the IP are presented in this section.

# 4.1 Overview of Product and Manufacturing Process for Clinical Trial Material

Novavax's Quad-NIV is based on purified, recombinant full-length HA that self-assembles into distinct nanoparticle structures of approximately 20 to 40 nm [Smith 2017]. The baculovirus/Spodoptera frugiperda (Sf9) insect cell system is used to clone and express recombinant influenza HAs from the influenza strains recommended for the 2019-20 Northern Hemisphere influenza season: A/Brisbane/02/2018 (H1N1) pdm09; A/Kansas/14/2017 (H3N2); B/Maryland/15/2016 (Victoria lineage); B/Phuket/3073/2013 (Yamagata lineage) [VRBPAC 2019, WHO 2019].

Matrix-M1 is a saponin-based adjuvant, which is co-administered with an antigen to induce an enhanced immune response. Matrix-M1 is manufactured by mixing defined, partially-purified extracts of the bark of the *Quillaja saponaria* Molina tree, termed Fraction-A and Fraction-C, with cholesterol and phosphatidylcholine in the presence of a detergent.

# 4.2 Manufacture of Bulk Antigen

# 4.2.1 Recombinant Baculovirus

The recombinant influenza HA genes are cloned into *E. coli* flashBAC GOLD baculovirus transfer vectors (Oxford Expression Technologies, Oxford, UK). The HA genes are under the transcriptional control of the baculovirus AcMNPV polyhedrin promoter at the 5' end and includes a poly (A) sequence at the 3' end. For each influenza strain, recombinant baculovirus expressing a HA gene are identified, plaque-purified, and amplified for use in the manufacture of recombinant influenza HA antigens.

#### 4.2.2 Production and Purification of Quad-NIV

Manufacture of each HA protein antigen is initiated by infecting Sf9 cells in exponential growth with baculovirus containing the strain-specific HA gene. After infection, cells are collected by centrifugation, washed with a detergent-free buffer, and then lysed in the presence of detergent to release membrane-bound HA protein. Leupeptin hemi-sulfate salt is added to the lysis buffer to protect the HA protein from cellular proteases released during the lysis step. The supernatant containing the HA protein is separated from cell debris through the use of depth filtration before it is purified on an ion exchange trimethylaminoethyl (TMAE) column. The flow-through fraction is then loaded onto a Capto Blue mixed-mode chromatography to capture and remove additional baculovirus and Sf9 host cell proteins, while HA is recovered in the flow-through fraction. Nanofiltration is then performed to remove viruses from the HA product stream. The HA protein is then loaded onto a lentil lectin column, which selectively binds the glycosylated protein. After washing, the HA protein is eluted from the column with buffer containing methyl-α-D-mannopyranoside (MMP) and polysorbate 80 (PS80). Eluted fractions are processed by tangential flow filtration, to concentrate the HA product and exchange it into the
final formulation buffer. The product is then diluted to a final formulation containing sodium phosphate and PS80, and then filtered (0.22 µm) to produce bulk drug substance that is clear and colorless, and contains no preservatives. Each HA bulk drug substance is stored at  $\leq$  -60°C until the 4 strains are mixed and diluted to the target concentration with buffer, and filled as drug product. The final composition of the drug product formulation is 25 mM sodium phosphate, 150 mM sodium chloride, 100 mM arginine hydrochloride, 5% w/v trehalose, and 0.03% PS80, pH 7.5.


#### 4.2.3 Manufacture of Matrix-M1 Adjuvant

Matrix-M1 is manufactured by mixing defined, partially-purified extracts of the bark of the Quillaja saponaria Molina tree, termed Fraction-A and Fraction-C, with cholesterol and phosphatidylcholine in the presence of a detergent. Detergent removal by diafiltration results in the formation of stable cage-like structures of 2 types, designated Matrix-A and Matrix-C, based on the precise Quillaja fraction incorporated. The designation, Matrix-M, refers generically to a blend of Matrix-A and Matrix-C particles together at any ratio. An 85:15 ratio (by weight) of Matrix-A and Matrix-C particles, respectively, yields Matrix-M1. For a more detailed description of the manufacturing process of Matrix-M1 adjuvant, refer to the current Matrix-M Adjuvant Safety Data Supplement.

#### 4.3 **Description of Clinical Trial Dosage Formulation**

Quad-NIV drug product co-formulated with Matrix-M1 adjuvant is filled directly into vials at appropriate concentrations. The buffer composition is the same as bulk antigen concentration alone, ie, 25 mM sodium phosphate, 150 mM sodium chloride, 100 mM arginine hydrochloride, 5% w/v trehalose, and 0.03% PS80, pH 7.5. The co-formulated drug product will be filled into 2R single-use glass vials.

#### 4.4 Fluzone Quadrivalent – Active Comparator

Fluzone Quadrivalent® (Sanofi Pasteur) will be administered based on manufacturer's instructions, which will be provided in the Pharmacy Manual.

#### 4.5 Investigational Product Packaging, Storage, and Handling

All IPs will be packaged in validated shipping containers for distribution to the investigational sites under refrigerated conditions. The vials and cartons will be labeled with the following information: manufacturer's name and address, product name, manufacture date, storage requirements (2 - 8°C), directions for use, and any other investigational product labeling appropriate to the jurisdiction in which the trial is conducted. Fluzone Quadrivalent will be packaged, shipped, and stored based on manufacturer's instructions. All IP and comparator materials should be stored at 2 - 8°C in a temperature-monitored refrigerator. Access to this refrigerator should be limited to designated site personnel.

#### 4.6 Compliance and Drug Accountability

All quantities of the test articles must be reconciled at the completion of enrollment and a written explanation provided for any discrepancies. Unless specific written instructions to the contrary are provided by Novavax, all unused test articles are to be inventoried, and either destroyed or returned to Novavax (or designee) by the clinical site upon notice by Novavax or the site monitor. All used vials will be accounted for on the clinical site's IP Dispensation Log by applying the tear-off portion of the vial/syringe label.

### 5 SELECTION OF TRIAL SUBJECTS

### 5.1 Inclusion Criteria

Subjects must meet all of the following criteria to be eligible to participate:

- 1) Clinically-stable adult male or female,  $\geq 65$  years of age. Subjects may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:
  - Ambulatory status, living independently in the community or in a residential facility providing minimal assistance (eg, meal preparation and transport),
  - Absence of changes in medical therapy within 1 month due to treatment failure or toxicity,
  - Absence of medical events qualifying as serious adverse events within the prior 2 months, and
  - Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the investigator.
- 2) Willing and able to give informed consent prior to trial enrollment, and
- 3) Living in the community and able to attend trial visits, comply with trial requirements, and provide timely, reliable, and complete reports of adverse events.

### 5.2 Exclusion Criteria

Subjects will be excluded if they meet any of the following criteria:

- 1) Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of study vaccination.
- 2) Participation in any previous Novavax's influenza vaccine clinical trial(s).
- 3) History of a serious reaction to prior influenza vaccination, known allergy to constituents of Fluzone Quadrivalent or polysorbate 80.
- 4) History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
- 5) Received any vaccine in the 4 weeks preceding the trial vaccination and any influenza vaccine within 6 months preceding the trial vaccination.
- 6) Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
- 7) Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.

- 8) Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the trial vaccine.
- 9) Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
- 10) Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
- 11) Known disturbance of coagulation.
- 12) Suspicion or recent history (within 1 year of planned vaccination) of alcohol or other substance abuse.

### 6 TRIAL ASSESSMENTS AND PROCEDURES

A trial schematic flowchart is provided in Appendix 1. A detailed description of procedures performed at each visit is provided in Section 6.1.

### 6.1 Trial Visit Procedures

### 6.1.1 Day 0 - Screening Visit

The following procedures will be performed on the day of the planned vaccination:

- Written informed consent will be obtained in conformance with Section 11.3 of this protocol.
- Inclusion and exclusion criteria review consistent with Section 5.
- Review of medical history, including influenza vaccination history in the previous 3 years (with emphasis on 2018-19 vaccine) and history of adverse reactions to prior influenza vaccines and allergies.
- Medication history, including concomitant medications and vaccines within the last year.
- Physical examination including the head, eyes, ears, nose, and throat (HEENT), abdomen, extremities, and at least inguinal, cervical, and axillary nodes, gross motor function, and skin; vital signs (heart rate, blood pressure, respiratory rate, and oral temperature); height and weight.

Note that further procedures may be performed at the investigator's discretion in order to adequately screen subjects against eligibility criteria and/or to confirm medical history. Potential subjects who meet all of the inclusion criteria and none of the exclusion criteria may be enrolled. Note: Subjects should be free of acute illness (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature  $\geq 38.0^{\circ}$ C) in order to receive the test article injection. Subjects presenting with an acute illness on Day 0 may return to the trial site within the next 7 days, as the enrollment timelines allow, to receive their injection provided symptoms have resolved.

# 6.1.2 Day 0 - Injection Visit

All subjects with confirmed eligibility will have the following procedures performed:

- Blood draw for baseline immunogenicity testing (20 mL, see Section 7.1).
- A subset of approximately 140 subjects from several pre-designated clinical sites (to target approximately 70 evaluable subjects per treatment group) will provide additional blood samples (27 mL per visit) at 4 time points (ie, Days 0, 7, 28, and 182) to support testing of cell-mediated immune responses (CMI). Note: All subjects at several pre-designated CMI testing sites will participate in CMI blood sampling and the Informed Consent document at those sites will be adjusted accordingly.
- Randomization to a treatment group.
- Alcohol swab cleansing of the injection site followed by IM injection of the assigned trial treatment into the deltoid muscle of the non-dominant arm. *Note: If the non-dominant arm*

is not available for the injection due to post-surgical changes, skin changes, or prior injury, the dominant arm may be used.

- Monitoring for any AEs for approximately 30 60 minutes following vaccination.
- Post-injection vital sign collection (heart rate, blood pressure, respiratory rate, and oral temperature) at 30 60 minutes following vaccination.
- Distribution of the subject diary, thermometer, and a measuring tool to facilitate documentation of any AEs (solicited and unsolicited), concomitant medications, physicians visits, or hospitalizations, occurring from the time of discharge from the trial clinic on Day 0 through Day 6 (inclusive). Subjects will also be instructed to call the trial clinic for any Grade 3 (severe) solicited or unsolicited health events, and/or health status changes of concern to the subject.
- Schedule the Day 7 or 28 visit before subjects may be dismissed from the clinic.

### 6.1.3 Day 3 (± 1 day) - Safety Telephone Contact

• Using an IRB-approved script, the trial staff will contact the subjects using a telephone call to query for any Grade 3 solicited or unsolicited event and/or SAE experienced, and any concomitant medications taken for these events since the last visit. Subjects may be asked to return to the clinic for an unscheduled visit to evaluate the event(s) at the trial investigator's discretion.

# 6.1.4 Day 7 (± 1 day) - Follow-up Visit

A subset of approximately 140 subjects who were enrolled at several pre-designated clinical sites, and who provided blood for CMI responses at Day 0, will return to the clinic on Day 7 for the following procedures:

- Vital sign collection (heart rate, blood pressure, respiratory rate, and oral temperature).
- Interval history to query for any unsolicited AEs, including MAEs, SNMCs, or SAEs, occurring since the last trial visit, and any concomitant medications taken. A directed physical examination may be performed at the investigator's discretion to evaluate any AEs.
- Blood draw to assess CMI responses (27 mL).
- Schedule the Day 28 visit.

### 6.1.5 Day 28 (± 4 days) – Follow-up Visit

All subjects will return to the clinic on approximately Day 28 for the following procedures:

- Vital sign collection (heart rate, blood pressure, respiratory rate, and oral temperature).
- Review and collection of subject diary.
- Blood draw for immunogenicity assessments (20 mL) for all subjects.
- Blood draw to assess CMI responses (27 mL) for a subset of approximately 140 subjects who were enrolled at several pre-designated clinical sites.

- Interval history to query for any unsolicited AEs, including MAEs, SNMCs, or SAEs, occurring since the last trial visit, and any concomitant medications taken. A directed physical examination may be performed at the investigator's discretion to evaluate any AEs.
- Schedule the Day 90 telephone contact and the Day 182 in-clinic visit.

## 6.1.6 Day 90 (± 7 days) - Safety Telephone Contact

• Using an IRB-approved script, the trial staff will contact the subjects using a telephone call to query for any MAEs, SAEs, and SNMCs since their last visit, and any concomitant medications taken for these events.

# 6.1.7 Day 182 (± 7 days) - Follow-up Visit

At Day 182, all subjects will return to the clinic for the following procedures:

- Vital sign collection (heart rate, blood pressure, respiratory rate, and oral temperature).
- Blood draw for immunogenicity assessments (20 mL) for all subjects.
- Blood draw to assess CMI responses (27 mL) for a subset of approximately 140 subjects who were enrolled at several pre-designated clinical sites.
- Interval history to query for any MAEs, SNMCs, or SAEs occurring since the last telephone contact, and any concomitant medications taken for these events. A directed physical examination may be performed at the investigator's discretion to evaluate any AEs.
- Schedule the end of the trial (Day 364) telephone contact.

# 6.1.8 Day 364 (± 14 days) – Safety Telephone Contact

- Using an IRB-approved script, the trial staff will contact the subjects using a telephone call to query for any MAEs, SAEs, and SNMCs since their last visit, and any concomitant medications taken for these events.
- This visit will mark the end of the trial for the subjects.

#### 6.2 Unscheduled Visits

Unscheduled visits are defined as any visits performed to the site outside of the regular visit schedule and can occur at the investigator's discretion for any other trial procedures deemed necessary. Subjects will be encouraged to notify the investigator if any severe (Grade 3) local or systemic solicited AEs occur within the 7-day post-dosing period (eg, from Day 0 through Day 6), or if any severe, serious, or otherwise concerning AEs occur at any time following dosing. If symptoms are presented that would require a physical exam to adequately assess potential AEs, the exam should be performed and vital signs collected.

# 6.3 Concomitant Therapy

Subjects may receive all concomitant medications and procedures deemed necessary to provide adequate healthcare during the trial, with the exception of those specified in the exclusion criteria. Routine medical standards of care are permitted, including vaccines needed for emergent indications (eg, tetanus booster in response to a penetrating injury). Routine (ie, non-emergent) vaccinations, except the seasonal influenza vaccine, are permitted for all

subjects after completion of the Day 28 trial visit. Subjects who receive a seasonal influenza vaccine outside of the study before Day 364 will be considered protocol deviations.

Concomitant medications, procedures, and hospitalizations will be recorded throughout the trial including the period from the day informed consent is obtained through the end of trial follow-up. All new or changed concomitant medications taken through Day 28 will be recorded; thereafter, only concomitant medications taken for MAEs, SNMCs, or SAEs will be recorded. The investigator will document the reason for use of the concomitant medication.

# 6.4 Declining Trial Treatments or Procedures

Subjects have the right to decline trial treatment or other trial procedures for any reason at any time during the trial. This trial contemplates one injection of either Quad-NIV with Matrix-M1 adjuvant or Fluzone Quadrivalent. Refusal of the investigational test article on Day 0 constitutes trial withdrawal without exposure, and no further follow-up is required. If a subject declines trial procedures subsequent to receipt of the investigational product, it should be recorded as a protocol deviation and the reason should be clearly documented in the source document. The subject will be asked to complete all other trial procedures as applicable. If the subject does not wish to remain in the trial, the subject can choose to withdraw consent and discontinue at any time as outlined in Section 6.5.

The investigator may, at his/her discretion, restrict a subject from receiving trial treatment or other trial procedures if he/she considers it to be in the subject's best interest to do so, but can suggest that the subject remain in the trial to be followed for safety if the subject has received a test article. In this situation, the reason for not performing the trial treatment and/or procedure should also be recorded as a protocol deviation and clearly documented in the source document.

### 6.5 Premature Discontinuation from Trial

Subjects who provide consent but are found to be ineligible on screening will be informed of the reason for ineligibility and may be provided with local medical referral by the investigator as appropriate, but will receive no further trial follow-up.

Subject participation in the trial is strictly voluntary. Subjects have the right to withdraw from the trial at any time and for any reason, without penalty. The investigator may also, at his/her discretion, discontinue subjects from the trial if he/she considers it to be in the participant's best interest to do so, or if the subject is not willing or able to comply with the trial requirements. Novavax will be notified immediately by the investigator if a subject prematurely ends trial participation. The reason for early discontinuation will be clearly documented in the electronic case report form (eCRF). A withdrawal due to an AE will initiate additional reporting requirements as outlined in Section 8.3.

In the event of early termination, investigators will make every reasonable effort to perform trial completion procedures. Trial completion procedures will include a query for any MAEs, SNMCs, or SAEs occurring since the last trial visit, and any concomitant medications taken to treat these events. If the subject discontinues from the trial prior to the Day 28 visit, sites will

request the subjects to provide blood samples for serology testing (20 mL). Subjects that terminate from the trial early will not be replaced.


#### 6.6 **Protocol Deviations**

A protocol deviation (PD) will be defined as a failure to comply with the requirements set forth in the protocol. PDs may be determined programmatically through the course of the trial. Examples of programmatically-determined PDs are provided in Table 2.

**Table 2: Programmatically-Determined Protocol Deviations** 

| Missed Visit |
|--------------------------|
| Out of Window Visit |
| Trial Procedure Not Done |
| Randomization Error |

#### 6.7 **Trial Termination**

Novavax reserves the right to terminate the trial at any time for any reason. If and when the trial is terminated (either prematurely or as scheduled), the investigator will notify the IRB for the trial and other authorities, as required by local regulatory requirements.

The scheduled end of the trial will be the completion of the last Day 364 follow-up visit with the last trial subject.

### 7 TRIAL LABORATORY REQUIREMENTS

Appendix 3 specifies the maximum amount of blood (up to 168 mL) to be drawn for immunogenicity laboratory assessments to be completed throughout the trial.

# 7.1 Serological Assessments of Immunogenicity

Immunogenicity assessments will be made on subject sera collected on Days 0, 28, and 182. The primary measure of immunogenicity for the trial is serum Day 28 HAI antibody titer specific for the HA receptor binding domains of each of the virus strains included in Quad-NIV using egg-propagated virus as the agglutinin in the HAI assay. The secondary measure of immunogenicity includes HAI titers specific for the HA receptor binding domains of vaccine-homologous and antigenically-drifted strains on Days 0 and 28 using both egg-propagated virus and VLP as the agglutinin in the HAI assay; an additional time-point at Day 182 may also be tested. In addition, neutralizing antibody titers specific for the virus strains included in Quad-NIV, as well as selected antigenically-drifted strains, may be evaluated.

# 7.1.1 Hemagglutination Inhibition (HAI) Assay

# 7.1.1.1 Egg-Propagated HAI

Briefly, sera will be treated with receptor-destroying enzyme (RDE) to remove non-specific inhibitors of hemagglutination, followed by heat-inactivation, and then plated into microtiter wells, starting with an initial dilution of 1:10 and followed by a series of 2-fold dilutions. The HA antigen (ie, egg-propagated whole virus) and human erythrocyte suspension will be added to designated wells in 2 steps, with mixing and incubation at each step. The titration endpoint will be taken as the highest dilution that demonstrates complete inhibition of hemagglutination. The serum HAI titer will be calculated from the GMT of duplicate test results. The HAI assay, as described in P\_SOP\_02076, will be validated for this Phase 3 trial in Novavax Clinical Immunology Laboratory under the supervision of Dr. Joyce Plested, Senior Director of Clinical Immunology.

#### 7.1.1.2 VLP-based HAI

Due to the documented inability of recent A(H3N2) strains to agglutinate avian or small mammal red blood cell reagents in hemagglutination inhibition (HAI) assays and, in addition, the presence of immunologically-significant mutations induced by egg passage in the HA of these strains [Zost 2017], vaccine immunogenicity will be assessed by the classical HAI method adapted with 140 - 190 nm recombinant wild-type hemagglutinin virus-like particles (HA-VLPs), reflecting the amino acid sequence of circulating virus, as the agglutinating agent and human type-O red blood cells (RBCs) as the agglutination target in order to restore assessment of HAI antibody activity. Briefly, sera will be first treated with RDE to remove non-specific inhibitors of hemagglutination, followed by heat-inactivation, and then plated into microtiter wells, starting with an initial dilution of 1:10 and followed by a series of 2-fold dilutions. The HA-VLPs and human erythrocyte suspension will be added to designated wells in 2 steps, with mixing and incubation at each step. The titration endpoint will be taken as the highest dilution that demonstrates complete inhibition of hemagglutination. The serum HAI titer will be calculated from the GMT of duplicate test results. The HAI assay will be validated

for this Phase 3 trial and performed as described in P\_SOP\_02041 in Novavax Clinical Immunology Laboratory under the supervision of Dr. Joyce Plested, Senior Director of Clinical Immunology.


#### **Microneutralization Assay** 7.1.2

The influenza virus microneutralization assay will be based on the WHO manual for the laboratory diagnosis and virological surveillance of influenza, with minor modifications [WHO 2011]. Briefly, subject test sera will be heat-inactivated at 56°C for 30 minutes. Sera will be prepared in 3-fold serial dilutions (starting from 1:10) in duplicate, in 96-well plates. Positive and negative serum controls will also be included. An approximate tissue culture infective dose of 100 (TCID<sub>50</sub>) wild-type cell-derived virus will be added and incubated for 120 minutes at  $37^{\circ}\text{C} \pm 2^{\circ}\text{C}$  in  $5.0\% \pm 1\%$  carbon dioxide (CO<sub>2</sub>) for influenza A virus and at  $32^{\circ}\text{C} \pm 2^{\circ}\text{C}$  in 5.0% ± 1% carbon dioxide (CO<sub>2</sub>) for influenza B virus. After incubation, 100 μL of trypsinized Madin Darby Canine Kidney (MDCK) cells at a concentration of 1.5 x 10<sup>5</sup>/mL will be added to each well and incubated for 18 to 22 hours at  $37^{\circ}\text{C} \pm 2^{\circ}\text{C}$  in  $5.0\% \pm 1\%$  CO<sub>2</sub> for influenza A virus and at  $32^{\circ}$ C  $\pm 2^{\circ}$ C in  $5.0\% \pm 1\%$  carbon dioxide (CO<sub>2</sub>) for influenza B virus. On Day 2, plates will be fixed, blocked, and incubated with mouse anti-influenza A nucleoprotein (NP) monoclonal antibody blend (MAB8251 for influenza A viruses or MAB8661 for influenza B viruses, EMD Millipore, Temecula, CA), followed by washing and incubation with a peroxidase-conjugated goat anti-mouse immunoglobulin G (IgG, Kirkegaard and Perry Laboratories, Gaithersburg, MD). Finally, plates will be washed and incubated with 3,3',5,5'-tetramethylbenzidine substrate (Sigma) and the optical density (OD) will be read after adding the stop solution. A sample titration curve is plotted OD against dilution using a 4-parameter curve fit. The sample neutralizing titer is interpolated on the titration curve as reciprocal of dilution at the OD that 50% of MDCK cells are infected. A 4-parameter fit (SoftMax Pro software) will use the following equation to determine the OD value at which 50% of the MDCK cells are infected:

X = [(average OD of virus control wells) + (average OD of cell control wells)] / 2

The microneutralization assay (Novavax P\_SOP\_02069) will be qualified before use and will be performed in the Novavax Clinical Immunology Laboratory under the supervision of Dr. Joyce Plested, Senior Director of Clinical Immunology.

#### 7.2 Assessments of Cell-Mediated Immunity

#### Assessment of T Cell Responses Based on Intracellular Cytokine 7.2.1 Staining

Human PBMCs are cultured in 96-well U-bottom plates at a density of 1 x 10<sup>6</sup> cells/well and treated with anti-CD28 and anti-CD49d antibodies. At the same time, the samples will be treated with HA protein from the tested strains or a heterologous strain, a positive control for T cell activation, or medium only (negative control). After incubation at 37°C for 6 hours in the presence of BD GolgiPlug<sup>TM</sup> and BD GolgiStop<sup>TM</sup> (BD Biosciences) for the last 4 hours, cells are labelled for surface markers (CD3, CD4, CD8, CD45RA, and CCR7 [BD Biosciences, San Jose, CA]) and the LIVE/DEAD® indicator dve (Life Technologies, NY) is added. The

qNIV-E-301 Protocol Page 48

intracellular cytokines are detected by antibodies specific for IFN- $\gamma$ , TNF- $\alpha$ , and IL-2. Expression of CD40L will also be tested. The samples are processed using a LSR-Fortessa flow cytometer (Becton Dickinson, San Jose, CA). Data are analyzed using Flowjo software version 10 (Tree Star Inc., Ashland, OR). A limited qualification of this assay will be performed prior to its use in clinical testing.

# 7.2.2 Assessment of Memory B Cell Response Based on Elispot Analysis.

HA-specific memory B cells are tested using Elispot analysis. PBMCs are cultured in the presence of R848 and human IL-2 for 5 days, and then added into plates that were pre-coated with Flu HA proteins of the tested strains. Flu HA-specific antibody-secreting cells are detected and counted by HRP conjugated anti-human IgG antibody.

# 7.3 Retention and Use of Archived Specimens

Subject serum samples may be archived by Novavax or its contractors for a period not to exceed 25 years. Archived samples may be used for repetition of the assays listed in Section 7.1 using different influenza antigens, or for other exploratory assays of influenza virus immunity or vaccine response in development. Archived sera may also be used for clinical laboratory testing for safety if needed to evaluate an adverse event, provided that a) sample storage falls within conditions previously validated by the clinical laboratory to yield interpretable results (or an appropriate control strategy can be used to evaluate potential storage impacts), and b) such testing will not include either assays to detect human immunodeficiency virus (HIV) infection, or any human genetic testing. Archived serum samples may also be used to create positive or negative panels for quality control or for assay development related to influenza virus or other infectious diseases (excluding HIV), in which case they will be anonymized.

### 8 TRIAL ASSESSMENT OF SAFETY

### 8.1 Adverse Events

Adverse events (AEs) are defined as any unfavorable or unintended change in the physical, psychological, or biochemical condition of the subject. An AE temporally related to participation in the trial or due to a procedure performed in the trial, will be documented whether or not considered related to the test article. This definition includes intercurrent illnesses and injuries, and exacerbations of pre-existing conditions. Stable pre-existing conditions which do not change in nature or severity during the trial are not considered AEs; however, these should be collected as part of the medical history. AEs will be considered treatment emergent from the date and time of the first administration of the investigational product.

Data concerning all classes of adverse events will be collected at scheduled visits from the time informed consent is obtained on Day 0 through Day 28, inclusive. After these specified days, data concerning MAEs, SNMCs, and SAEs will be collected (see Sections 8.1.4 and 8.2 for details of these AEs), as well as additional information regarding outcomes/resolutions of AEs reported prior that had no stop date recorded. In addition to the scheduled visits, subjects will be instructed to notify the investigator and/or return to the clinic if any severe AE (solicited or otherwise) or event fulfilling the definition of an SAE occurs at any time following vaccination. If at a scheduled or unscheduled visit, symptoms are presented that would require a physical exam to adequately assess potential AEs, the exam should be performed and vital signs collected. Adverse events will be recorded as observed by the investigator, designated personnel, or as provided by the subject on the diary card or during the in-person visit. Full details of the AE (ie, nature, date of onset, and recovery, as well as an assessment of severity, relationship to trial treatment [unsolicited events only], seriousness, treatment, and outcome) will be recorded in the source documentation and captured in the eCRF, and will generally require the investigator(s) causality assessment, except as discussed below.

# 8.1.1 Solicited Adverse Events/Subject Diary

Subjects will be provided with a diary for the documentation of any AEs, daily recording of their body temperature and certain common post-vaccination symptoms, and concomitant medications and procedures starting on vaccination day and for 6 days following the Day 0 vaccination (ie, from Day 0 through Day 6, inclusive). A series of local injection site and systemic reactions that are reasonably likely to occur in vaccine programs (Table 3) will be solicited daily in the diary and standardized severity grades offered to the subject. Subjects will report injection site events occurring on the deltoid where the test article was administered. A standard tool for the measurement of visible local reactions will be provided (see example provided in Appendix 1) as will a digital oral thermometer. Subjects will also be asked to record any physician visits or hospitalizations, and any unsolicited AEs experienced during Day 0 through Day 6. In addition to reporting Grade 3 solicited adverse events in the diary card, subjects should be encouraged to contact the investigator by telephone if these occur. The investigator may request an *ad hoc* clinic visit at his/her judgment, and should enter any Grade 3 solicited adverse events reported by telephone in the eCRF promptly, even if the balance of diary data is not yet available.

**Table 3: Listing of Diary Solicited Events** 

| Injection Site | | Systemic Even | nts |
|---|---|---|---|
| (Local) Events: | General | Gastrointestinal | Respiratory/Facial |
| Pain | Oral temperature | Nausea | Eye redness |
| Bruising | Chills | Vomiting | Facial swelling |
| Redness | Muscle pain | Diarrhea | Eyelid swelling |
| Swelling | Joint pain | | Hoarseness |
| | Headache | | Sore throat |
| | Fatigue | | Cough |
| | | | Difficulty breathing |
| | | | Wheezing |
| | | | Chest tightness |
| | | | Difficulty swallowing |

Note: All events listed will be solicited by diary for 7 days post-dosing. Subjects will report injection site events occurring on the arm where the test article was administered. Events reported outside the solicitation window will be categorized and reported as unsolicited AEs.

Standard severity grading definitions will be provided in the diary. Grading of visible, measurable injection site reactions will be based on the Food and Drug Administration (FDA) Guidance for Industry, Toxicity Grading Scale (TGS) for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007). Definitions are summarized in Table 5. Oral temperatures will be collected as a continuous variable and graded by the investigator based on ranges provided in the TGS as shown in Table 6.

Investigators will not be required to assess causality of solicited adverse events specifically named in the diary if onset is during the solicitation period (these will be presumed to be treatment-related). Adverse events consistent with the solicited adverse events listed in the diary, but with onset after the solicitation period (ie, Day 7 thereafter), will be captured as unsolicited AEs and are subject to all procedures for unsolicited AE data.

Solicited AEs, collected from the subject diary, which continue after the collection period (ie, on or after Day 7 for vaccination-emergent events) will be followed to resolution. The continuing, solicited AE will be captured by verbatim term on an "AE eCRF" page. The investigators will be required to assess severity of the continuing solicited adverse event(s) starting from the time after the last diary entry until resolution.

#### 8.1.2 Unsolicited Adverse Events

Any AEs reported spontaneously by subjects will be categorized as unsolicited events and Medical Dictionary for Regulatory Activities (MedDRA) coded by system organ class (SOC) and preferred term (PT). Solicited events with an onset after the solicitation period will also be classified as unsolicited AEs. Unsolicited events that occur within 7 days following vaccination should also be recorded in the subject diary. If any Grade 3 unsolicited event is reported during this period, subjects should be encouraged to contact the investigator by telephone. The investigator may request an *ad hoc* clinic visit at his/her judgment, and should enter any Grade 3 unsolicited adverse event reported by telephone in the unsolicited AE eCRF promptly, even if the balance of diary data is not yet available. All unsolicited AEs will be assessed for severity

(as defined in Section 8.1.2) and for causality (as discussed in Section 8.5), and will be documented in the source documents and captured in the eCRF.

### 8.1.3 Vital Sign Abnormalities as Adverse Events

For purposes of reporting vital sign abnormalities as AEs, those values that show an increase in the toxicity grade relative to the baseline values (in the same subject) and *attain* at least a Grade 2 (eg, normal or Grade 1 to Grade 2, or Grade 2 to Grade 3) should be reported as an AE, at the investigator's judgement. Investigators may report lesser abnormalities as AEs if indicated based on clinical judgment. Abnormal vital signs may be repeated at the investigator's discretion, and because these measures are highly labile, should only be reported as AEs when the investigator believes there is a persistent and meaningful and clinically-significant physiologic change. If multiple assessments of vital signs are made, then only the most recent measurement will be reported. Vital sign abnormalities which are the logical consequence of another diagnosis (eg, irregular tachycardia in a subject with atrial fibrillation or fever in a subject with pneumonia) need not be reported separately.

# 8.1.4 Medically-attended Events and Significant New Medical Conditions

These classes of events will be collected at all trial visits, and if offered spontaneously by the subject at any time.

Medically-attended events (MAEs) are adverse events which result in an unscheduled visit to a healthcare provider due to symptomatic illness or injury. These may include office visits, clinic visits, home consultations, or emergency room evaluations for non-life-threatening events that do not result in hospitalization (life-threatening events or hospitalizations are SAEs, see Section 8.2).

Significant new medical conditions (SNMCs) are adverse events that are new (that is, not present at baseline), clinically significant (meaning that they imply an important change in the subject's long-term health status), and typically chronic (requiring an ongoing change in the subject's medical management). This category is not meant to include minor or transient diagnoses or age-related changes. For example, while new diagnoses of presbyopia or tinea versicolor are chronic conditions, they are not SNMCs because no significant change in health status is implied. Similarly, adverse events which are isolated, treatable events that resolve and do not require chronic therapy are also not SNMCs (examples could include an uncomplicated acute urinary tract infection or a simple fracture resolved with conservative treatment and with no residual disability). In contrast, new diagnoses of rheumatoid arthritis or coronary artery disease are SNMCs because they imply a long-term change in health status and require ongoing medical management. Additionally, because it has been hypothesized that immunizations with or without adjuvant may be associated with autoimmunity, regulatory authorities have requested that Novavax instruct investigators to be especially vigilant regarding the AESIs listed in Table 4. Note that this regulatory request is not specific to Novavax's Quad-NIV or Matrix-M1 adjuvant; and there is no current evidence to suggest that the trial drugs in this protocol are, or are not, associated with these illnesses. The list is not intended to be exhaustive, nor does it exclude the possibility that other diagnoses may be AESIs.

**Table 4: Adverse Events of Special Interest** 

| Categories | Diagnoses (as MedDRA® Preferred Terms) |
|---|---|
| Neuroinflammatory Disorders: | Acute disseminated encephalomyelitis (including site specific variants: eg, non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis), cranial nerve disorders including paralyses/paresis (eg, Bell's palsy), Guillain-Barre syndrome (including Miller Fisher syndrome and other variants), immune-mediated peripheral neuropathies and plexopathies (including chronic inflammatory demyelinating polyneuropathy, multifocal motor neuropathy and polyneuropathies associated with monoclonal gammopathy), myasthenia gravis, multiple sclerosis, narcolepsy, optic neuritis, transverse myelitis, uveitis |
| Musculoskeletal and Connective Tissue Disorders: | Antisynthetase syndrome, dermatomyositis, juvenile chronic arthritis (including Still's disease), mixed connective tissue disorder, polymyalgia rheumatic, polymyositis, psoriatic arthropathy, relapsing polychondritis, rheumatoid arthritis, scleroderma (including diffuse systemic form and CREST syndrome), spondyloarthritis (including ankylosing spondylitis, reactive arthritis [Reiter's Syndrome] and undifferentiated spondyloarthritis), systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome |
| Vasculidities: | Large vessels vasculitis (including giant cell arteritis such as Takayasu's arteritis and temporal arteritis), medium sized and/or small vessels vasculitis (including polyarteritis nodosa, Kawasaki's disease, microscopic polyangiitis, Wegener's granulomatosis, Churg–Strauss syndrome [allergic granulomatous angiitis], Buerger's disease [thromboangiitis obliterans], necrotizing vasculitis and anti-neutrophil cytoplasmic antibody [ANCA] positive vasculitis [type unspecified], Henoch-Schonlein purpura, Behcet's syndrome, leukocytoclastic vasculitis) |
| Gastrointestinal Disorders: | Crohn's disease, celiac disease, ulcerative colitis, ulcerative proctitis |
| Hepatic Disorders: | Autoimmune hepatitis, autoimmune cholangitis, primary sclerosing cholangitis, primary biliary cirrhosis |
| Renal Disorders: | Autoimmune glomerulonephritis (including IgA nephropathy, glomerulonephritis rapidly progressive, membranous glomerulonephritis, membranoproliferative glomerulonephritis, and mesangioproliferative glomerulonephritis |
| Cardiac Disorders: | Autoimmune myocarditis/cardiomyopathy |
| Skin Disorders: | Alopecia areata, psoriasis, vitiligo, Raynaud's phenomenon, erythema nodosum, autoimmune bullous skin diseases (including pemphigus, pemphigoid and dermatitis herpetiformis), cutaneous lupus erythematosus, morphoea, lichen planus, Stevens-Johnson syndrome, Sweet's syndrome |
| Hematologic Disorders: | Autoimmune hemolytic anemia, autoimmune thrombocytopenia, antiphospholipid syndrome |
| Metabolic Disorders: | Autoimmune thyroiditis, Grave's or Basedow's disease, Hashimoto thyroiditis, diabetes mellitus type 1, Addison's disease |

**Table 4: Adverse Events of Special Interest** 

| Categories | Diagnoses (as MedDRA® Preferred Terms) |
|---|---|
| Other Disorders: | Goodpasture syndrome, idiopathic pulmonary fibrosis, sarcoidosis, pernicious anemia |

The eCRF will provide a field in which the investigator may designate AEs as MAEs, SNMCs, or both. Because of the significance of the designation for the subject's health, long-term medical management, and for evaluation of vaccine safety, SNMCs are expected to be substantiated diagnoses, not isolated symptoms which might or might not be a SNMC, and the investigator should record sufficient data in the eCRF to support the diagnosis.

#### 8.2 Serious Adverse Events

A SAE is defined as an AE that results in any of the following outcomes:

- Death,
- An immediate threat to life,
- In-patient hospitalization or prolongation of an existing hospitalization. (Hospitalization is defined as an actual admission, not a 24-hour stay or emergency room visit; note that elective surgeries, undertaken for conditions present prior to receipt of trial drug and without complication, should not be considered SAEs),
- A persistent or significant disability/incapacity (substantial disruption of an ability to conduct normal life functions), or
- A congenital anomaly or birth defect (not relevant to this protocol).

An important medical event that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias, or convulsions that do not result in in-patient hospitalization. Events which could have led to the above outcomes had they occurred with greater severity are not SAEs, but should be reported as AEs, MAEs, or SNMCs, as appropriate.

The eCRF will provide a field for designating an AE as an SAE. SAEs are associated with enhanced reporting requirements (see Section 8.3).

# 8.3 Safety Reporting Requirements and Timelines for SAEs and Certain Other Events

Any SAE must be reported (using the SAE Report Form) to Novavax Product Safety within 24 hours of the investigator's first knowledge of the event, regardless of the presumed relationship to the investigational product. The investigator or qualified designee must complete the SAE Report Form, sign, and transmit the completed form to Novavax Product Safety.

Initial reports of SAEs may be reported via fax or e-mail. Initial reports **must** be signed (physically or electronically) by the investigator or a qualified sub-investigator and transmitted to Novavax Product Safety **within 24 hours** of site awareness. When additional follow-up information becomes available, a written follow-up SAE Report Form must be completed, signed by the investigator or a qualified sub-investigator, and transmitted as soon as possible. The investigator is responsible for obtaining detailed information to support all SAE reports, including records of inpatient and outpatient care, laboratory reports, and autopsy or medical examiner reports.

The following events must also be reported to the Medical Monitor within 24 hours of the investigator's first knowledge of the event:

- Any withdrawal of consent after dosing due to an AE.
- Overdose (of a test article as specified in the protocol with or without an AE).
- Inadvertent or accidental exposure to the test article with or without an AE.
- Medication error (includes the administration of an incorrect treatment, an expired test article, a test article that has deviated from its required storage or refrigeration requirements, or any test article prior to documentation of informed consent).

Novavax will be responsible for notifications of SAEs to the relevant regulatory authorities; investigators will be responsible for IRB notification.

# 8.4 Severity

All AEs will be assigned severity by the subject and/or investigator (as applicable) according to the TGS. Subjects will also be able to indicate severity for any AEs experienced and record this in their diary according to the same scale. For quick reference, an abbreviated grading scale is provided in Table 5 for visible and non-visible local AEs and for systemic AEs for which severity is based on interference with daily activities and not numeric ranges, and in Table 6 for fever and gastrointestinal adverse events of nausea, vomiting, and diarrhea.

The severity of visually-evaluated local AEs will be a function of size. During the diary period, subjects will monitor the size of visible local AEs at the injection site using the Subject Measurement Tool (Appendix 4) which has concentric circles that correspond to the diameters specified in Table 5. For the purposes of reporting during the solicitation period (ie, Day 0 through 6) the subjects' observations will form the primary data. During clinic visits, investigators may measure any persisting local AEs with a ruler, documenting the size of the reaction at its widest diameter, using the numeric scale provided in Table 5 to assess for severity.

Non-visible local AEs (eg, pain) will be assigned a severity based primarily on interference with daily activities.

Systemic solicited AEs and unsolicited AEs will be assigned a severity grade based primarily on disruption of normal daily activities, with the exception of fever and select solicited gastrointestinal AEs that have their own distinct toxicity grades (Table 6). Medical care-seeking is typically absent for Grade 1 (mild) and often present for Grade 3 (severe) events, but is not the primary determinant of severity, since individuals behave differently in this regard.

Severity of vital sign abnormalities (including oral temperature, which is captured as a continuous variable) will be graded based on established ranges provided in the TGS and reported as an AE using the criteria outlined in Section 8.1.3.

**Table 5: Definition of Severity Grading for Adverse Events** 

| | Definitions for Lo | cal Adverse Events | Definitions for Systemic Adverse<br>Events |
|---|---|---|---|
| Severity<br>Grade | Visual Local AE Size Grading Description | Non-Visual Local AE<br>Grading Description | Systemic AE Grading Description |
| 0 – Normal | Reaction size<br>(greatest single diameter)<br>< 2.5 cm | No noticeable symptom | No noticeable symptom or finding |
| 1 – Mild | Reaction size<br>(greatest single diameter)<br>2.5 to 5.0 cm | Discomfort or tenderness<br>noticeable, but does not<br>interfere with normal<br>daily activities | Mild symptoms or diagnostic observations; intervention not indicated; no interference with normal activity |
| 2 – Moderate | Reaction size (greatest single diameter) > 5.0 to 10.0 cm | Moderate discomfort or<br>tenderness on firm<br>pressure; causes some<br>limitation of normal daily<br>activities | Moderate symptoms or diagnostic observations; some interference with normal activity, not requiring medical intervention |
| 3 – Severe | Reaction size<br>(greatest single diameter)<br>> 10.0 cm | Severe pain at rest, pain<br>or tenderness<br>immobilizes the injected<br>limb and prevents normal<br>daily activities | Severe symptoms, significantly<br>disrupts or prevents normal daily<br>activities, generally requires medical<br>attention/intervention |

Table 6: Severity Grade Definitions for Solicited Gastrointestinal Adverse Events and Fever

| | Gast | | | |
|---|---|---|---|---|
| Severity Grade | Nausea | Vomiting | Diarrhea | Fever |
| 0 – Normal | No noticeable symptom | No noticeable symptom | No noticeable symptom | < 38.0 |
| 1 – Mild | No interference<br>with activity, or 1<br>to 2 episodes/<br>24-hour period | No interference<br>with activity, or 1<br>to 2 episodes/<br>24-hour period | 1 to 3 unformed<br>(loose)<br>stools/24-hour<br>period | 38.0 to 38.4 |
| 2 – Moderate | Some interference with activity, or > 2 episodes/ 24-hour period | Some interference with activity, or > 2 episodes/ 24-hour period | 4 to 5 unformed<br>(loose)<br>stools/24-hour<br>period | 38.5 to 38.9 |
| 3 – Severe | Prevents daily<br>activity, or requires<br>intravenous<br>hydration | Prevents daily<br>activity, or requires<br>intravenous<br>hydration | ≥ 6 loose<br>stools/24-hour<br>period, or requires | > 38.9 |

Table 6: Severity Grade Definitions for Solicited Gastrointestinal Adverse Events and Fever

| | Gast | | | |
|----------------|--------|----------|-------------|-------|
| Severity Grade | Nausea | Vomiting | Diarrhea | Fever |
| | | | intravenous | |
| | | | hydration | |

# 8.5 Relationship (Causality)

The relationship of an AE to the test article must be assessed and documented by the investigator or a qualified sub-investigator. Based on the criteria described below, the investigator must classify the AE according to the following categories shown in Table 7.

**Table 7: Definition of Relationship for Adverse Events** 

| Relationship | Relationship Description |
|---|---|
| Unrelated / Unlikely | May or may not follow a reasonable temporal sequence from administration of the test article; |
| | No plausible mechanism based on known or suspected actions of the test article or product class; |
| | Readily explained by known characteristics of the subject's clinical state, common intercurrent illnesses, or other treatments administered to the subject. |
| Possibly | Follows a reasonable temporal sequence from administration of the test article; |
| | Based on known or suspected actions of the test article or product class, a plausible mechanism could exist; |
| | • May be reasonably explained by known characteristics of the subject's clinical state, common intercurrent illnesses, or other treatments administered to the subject; but the investigator deems this less likely than test article effect. |
| Probably | Follows a reasonable temporal sequence from administration of the test article; |
| | Based on known or suspected actions of the test article or product class, a plausible mechanism could exist; |
| | • Cannot be reasonably explained by known characteristics of the subject's clinical state, common intercurrent illnesses, or other treatments administered to the subject. |
| Definitely | Follows a reasonable temporal sequence from administration of the test article; |
| | Consistent with known actions of the test article or product class; |
| | • Cannot be reasonably explained by known characteristics of the subject's clinical state, common intercurrent illnesses, or other treatments administered to the subject. |
| | May be confirmed by re-challenge (if applicable). |

### 9 TRIAL DATA MANAGEMENT

# 9.1 Recording and Collection of Data

Novavax will provide sites with source document templates for the recording and collection of subject data. Data will be entered into an electronic data capture (EDC) system by site staff. All EDC entries will be completed as soon as possible after the subject's visit. Corrections to data in the EDC system will be documented in the electronic audit trail that is compliant to US FDA regulations (21 Code of Federal Regulations Part 11). The investigator will review data resident in the EDC and indicate by electronic signature that, to his/her knowledge, the data are complete and accurate. If further changes are made after this, the investigator will need to again sign the Investigator Signature Page electronically. Designated source documents will be signed and dated by the appropriate trial personnel. The investigator must agree to ensure completion and maintenance of source documents for each subject participating in the trial.

# 9.2 Data Quality Assurance

All trial data will be entered by clinical trial site staff with trial-specific EDC training into a computerized data management system via EDC. Statistical analyses of data will only be performed after all clinical monitoring and data queries have been resolved.

# 9.3 Monitoring

Novavax, as the Sponsor of this trial, is responsible for ensuring the proper conduct of the trial, in accordance with the Declaration of Helsinki (Amended Fortaleza, Brazil, 2013) and Good Clinical Practices (GCP) including, but not limited to, protocol adherence and the validity of the data recorded in the database. For the purposes of this trial, Novavax may transfer responsibility for the clinical monitoring to a CRO who may monitor on-site or remotely. Novavax and/or CRO are responsible for ensuring that the site(s) prepare complete, accurate, legible, and well-organized clinical trial data. On-site monitoring inspections will be routinely performed in order to review data entry of source documentation directly captured on paper and transcribed into the system, to ensure protocol adherence, to assess site operational capabilities, and to perform other monitoring activities that cannot be performed remotely. In addition, clinical monitors will provide ongoing support to ensure the investigator's continued understanding of all applicable regulations concerning the clinical evaluation of the investigational vaccine, and the proper execution of the protocol, as well as the investigator's reporting responsibilities.

The clinical trial sites will be monitored periodically for database accuracy and completeness, adherence to the protocol, regulatory compliance, safety reporting, clinical trial material accountability, and the maintenance of comprehensive source documents. When data entry has been completed by the appropriate trial staff, source documents verified and monitored by Novavax and/or CRO representatives, and reviewed by the investigator, the investigator should sign and date the *Investigator Signature Page*.

# 9.4 Audit and Inspection

Novavax CQA reserves the option to develop a Quality Assurance plan to ensure the integrity of the conduct of the clinical trial. CQA visits may be performed during the trial and post-trial by Novavax CQA or other personnel authorized by Novavax. Regulatory authorities reserve the right to audit trial sites following submission of data in regulatory applications. By signing this protocol, the investigator acknowledges that these inspection procedures may take place and agrees to provide access to the required subject records and other trial documentation. Further, the investigator agrees to inform Novavax and the IRB immediately of any scheduled or unscheduled inspection by regulatory authorities.

# 9.5 Adherence to and Changes to the Protocol

Any change or addition to this protocol will only be made when a protocol amendment has been written, approved, and signed by Novavax and the investigator before the change or addition can be considered effective, unless immediate implementation of a change is necessary to ensure the safety of subjects. This amendment must also be submitted to the IRB for approval and, when necessary, regulatory authority approval before implementation. Protocol amendments may affect consent forms of current and future subjects. Novavax will clearly specify when a protocol amendment includes safety, procedural, and/or efficacy information that will require specific informed consent form (ICF) text changes.

# 9.6 Retention of Records

It is the responsibility of the investigator and trial staff to maintain a comprehensive and centralized filing system of all trial-related documentation, which is suitable for inspection at any time by Novavax, its designees, and regulatory agencies. These should minimally include:

- Subject files including the completed eCRF (based on output from clinical database) on compact disc (CD), supporting source documentation, and the informed consent and any other subject information.
- Trial files (essential documents and regulatory files) including the protocol with all amendments, the IB, safety and protocol deviations meeting IRB reportable criteria, copies of all regulatory documentation, and all correspondence with the IRB, regulatory authority, and Novavax.
- Pharmacy files including all investigational vaccine shipment, receipt, storage, dispensing, and accountability records, and pharmacy-related correspondence.

In addition to the eCRF, the investigator will maintain adequate records that fully document the progress of the trial. Copies of these trial records and related documents must be kept on file by the investigator for a period of no less than 15 years (or longer if mandated by relevant local regulations). ALL DOCUMENTATION AND MATERIAL PROVIDED BY NOVAVAX OR A NOVAVAX REPRESENTATIVE FOR THIS TRIAL (CASE REPORT FORMS, PROTOCOL, ETC) ARE TO BE RETAINED IN A SECURE PLACE AND TREATED AS CONFIDENTIAL MATERIAL.

### 10 TRIAL STATISTICAL CONSIDERATIONS

This section includes a brief description of the statistical analyses that will be performed in this trial.

# 10.1 Subject Populations

The following subject populations will be used in all analyses:

- Safety Population Includes all trial subjects that provide consent, are randomized, and receive the test article. The Safety Population will be used for all safety analyses; and will be analyzed as actually treated.
- Per-Protocol Population (PP) Includes all subjects in the Safety Population that received the assigned dose of the test article according to protocol, have HAI serology results for Day 0 and Day 28, and have no major protocol deviations affecting the primary immunogenicity outcomes as determined by Novavax prior to database lock and unblinding. The PP Population will be the primary population used for immunogenicity analyses.
- Intent-to-Treat (ITT) Population Includes all subjects in the Safety Population that provide any HAI serology data. The ITT Population will be the secondary population used for any immunogenicity analyses and will be analyzed according to treatment as randomized. Analysis using the ITT population will not be performed if it differs from the PP population by ≤ 5% of the subjects for each of the 2 treatment groups.

#### 10.2 General

Continuous variables will be presented by summary statistics (eg, mean and standard deviation [SD] for the non-immunogenicity endpoints; geometric means and their 95% CI for the immunogenicity endpoints). Categorical variables will be presented by frequency distributions (frequency counts and percentages for the non-immunogenicity endpoints; percentages and their 95% CIs for the immunogenicity endpoints).

# 10.3 Demographics and Protocol Compliance

Demographic parameters and other baseline characteristics (eg, age, sex, race, and ethnicity) will be summarized by treatment group for all subjects in the safety population. The number and description of protocol deviations will be summarized for all enrolled subjects who signed the ICF and were randomized in to the study.

# 10.4 Analyses Addressing Protocol Objectives

# 10.4.1 Analyses of Primary Objectives

### 10.4.1.1 Immunogenicity

The Per-Protocol (PP) population (ie, randomized subjects who received the assigned dose of the test article according to the protocol, have HAI serology results at Day 0 and Day 28, and have no major protocol deviations) will be the primary population for immunogenicity analysis. A separate intent-to-treat (ITT) population analysis will not be produced unless > 5% of at least

1 treatment group is excluded from the PP population. No missing data will be imputed. For GMTs and GMRs, titers reported below the lower limit of quantitation (LLOQ, ie, below the starting dilution of assay reported as "< 10") will be set to half that limit (ie, 10/2 = 5).


For purposes of determining non-inferiority (and exploratory superiority) in immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, for all Quad-NIV homologous influenza strains (2 influenza A and 2 influenza B strains) at 28 days post-vaccination, derived/calculated endpoints will include:

- Two-sided 95% CIs for the ratio of Day 28 post-vaccination GMTs between Quad-NIV and Fluzone Quadrivalent will be constructed using log normal distribution. The log<sub>10</sub> values will be used to construct a CI using the analysis of covariance (ANCOVA) with treatment group and baseline at Day 0 (adjusted for intergroup variation in baseline [pre-vaccination] titers) as the covariates under two-sided type I error rate of 0.05. No type I error rate adjustments will be made. The mean difference and the corresponding CI limits will then be exponentiated to obtain the ratio of GMT and the corresponding CI.
- Two-sided 95% CIs for the difference of the SCRs between Quad-NIV and Fluzone Quadrivalent will be based on the Newcombe hybrid score (METHOD = SCORE riskdiff-option for PROC FREQ in SAS).

# 10.4.2 Analysis of Secondary and Exploratory Immunogenicity Objectives

Immunogenicity of 240 µg Quad-NIV co-formulated with 75 µg Matrix-M1 adjuvant, relative to a US-licensed comparator, Fluzone Quadrivalent, based on HAIs (assayed with both egg-propagated virus and wild-type VLP reagents) for all vaccine-homologous influenza A and B strains, and at least 1 antigenically-drifted A or B strain at Day 28 post-vaccination, will be measured in terms of:

- Geometric mean titer (GMT) defined as the antilog of the mean of the log-transformed HAI titers, on Days 0 and 28.
- Geometric mean ratio (GMR) defined as the ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs (GMR<sub>Post/Pre</sub>) on Day 28.
- Seroconversion rate (SCR) defined as proportion of subjects in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer  $\geq$  40, or a baseline reciprocal (Day 0) titer of  $\geq$  10 and a post-vaccination titer  $\geq$  4-fold higher on Day 28.
- Seroprotection rate (SPR) defined as the proportion of subjects with a reciprocal HAI titer  $\geq$  40 on Day 28.
- Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).

An additional time-point at Day 182 may also be tested.

Microneutralization (MN) responses at Days 0 and 28 post-vaccination will include:

- GMT defined as the antilog of the mean of the log-transformed neutralizing titer for a given treatment group.
- GMR defined as the ratio of post-vaccination and pre-vaccination neutralizing GMTs within the same treatment group (designated as GMR<sub>Post/Pre</sub>).
- SCR defined as proportion of subjects in a given treatment group with either a baseline reciprocal titer of < lower limit of quantitation (LLOQ) and a post-vaccination reciprocal titer 4-fold higher than the LLOQ, or a baseline reciprocal titer of ≥ LLOQ and a post-vaccination reciprocal titer ≥ 4-fold higher than the baseline titer.
- Ratio of GMTs between treatment arms at Day 28 post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).

An additional time-point at Day 182 may also be tested.

Analysis of exploratory CMI response endpoints will be performed on a subset of approximately 140 subjects from several pre-designated clinical sites (70 subjects per treatment arm) and results may be reported as an addendum to the main clinical study report.

# 10.4.3 Analyses Concerning Safety Objectives

Safety analysis will be descriptive and based on the safety population, defined as all subjects who received a dose of trial treatment. Safety will be summarized overall and by individual treatment arms based on solicited short-term reactogenicity post-injection on Day 0 - 6, 28-day all AE profile by MedDRA preferred term, and 1-year MAE, SAE, and SNMC profiles post-injection on Day 0. All AEs, including MAEs, SAEs, and SNMCs will be tabulated by severity, related (possibly, probably, or definitely vs non-related per investigator assessment), and severe and related. The number and percentage (with 95% CI) of subjects in each treatment group with a given term will be summarized. A listing and narratives of SAEs will also be produced.

# 10.5 Sample Size Considerations

This study has a single comparison between Quad-NIV and Fluzone Quadrivalent at Day 28 post-vaccination for the primary immunogenicity objective. No adjustment of the Type I error rate for multiple comparisons is warranted since the simultaneous successes of all 8 comparisons planned for the 4 strains contained in the vaccines and the two endpoints (GMT and SCR) are required for the demonstration of the primary non-inferiority objective of the study.

Non-inferiority is defined as the lower bound of the 2-sided 95% CI on the ratio of GMTs (Quad-NIV vs Fluzone)  $\geq 0.67$  (ie, unadjusted 1-sided p-value < 0.025 against the null hypothesis of H0: Ratio of GMT < 0.67) and the lower bound of the two-sided 95% CI on the difference of the SCRs (Quad-NIV - Fluzone)  $\geq$  -10% (ie, unadjusted 1-sided p-value < 0.025 against the null hypothesis of H0: Difference of SCRs < -10%).

For the calculation of sample size estimation, we used assumptions of true differences, ie, the ratio of GMTs (Quad-NIV vs Fluzone Quadrivalent) is 1.0 for all 4 homologous strains, and

the difference of the SCRs is -2% for each of the 4 homologous strains, based on the average performance in the previous trial (qNIV-E-201). To achieve an overall 90% power (ie, ~ 97.5% power for each of the 4 strains) to demonstrate a non-inferiority margin for SCR difference of -10%, the SCR of reference group (Fluzone Quadrivalent) is assumed to be 0.5 and the SCR of treatment group (Quad-NIV) is assumed to be 0.48 under the null hypothesis of inferiority (H0: Difference of SCRs < -10%). The significance level of the testing is 0.025. Sample size was estimated to be 1195 in each group by assuming equal size in each group. The sample size accounted for a 10% attrition rate for the per-protocol population such that the primary analysis population for all immunogenicity endpoints will be 1325 in each group.

In a previous trial (qNIV-E-201), the observed vaccine-homologous strain-specific standard deviations of  $\log_{10}$  HAI titers ranged from approximately 0.3 (B/Colorado/06/2017 and B/Phuket/3073/2013) to approximately 0.4 (A/Singapore/INFIMH-16-0019/2016 and A/Michigan/45/2015). The calculated power for each strain, unadjusted for multiple comparisons, is close to 100% to detect a 1.5-fold difference in GMTs. For 4 strains, this study is designed to exclude a GMT ratio of < 0.67 with 100% power. Therefore, for demonstrating non-inferiority for 4 strains with the true ratio of GMTs of 1.0 and the true SCR differences of -2%, this study provides  $\geq$  90% overall power.

For safety endpoints, the probability of observing at least 1 adverse event among 1325 subjects for Quad-NIV is > 90% if the true rate of such events is 0.18%. With 1325 subjects for Quad-NIV, observing no adverse events of interest (eg, vaccine-related SAE) would represent an upper bound of the 1-sided 95% CI on the percentage of such event is 0.2%.

# 10.6 Plan for Statistical Summaries and Analyses

# 10.6.1 Day 28 Unblinded Data Review

An unblinded data review will be conducted upon completion of Day 28 visits, which will include all primary endpoints (HAI antibody responses assayed with egg-propagated virus) testing of associated Day 28 serum samples for all 4 vaccine homologous influenza strains (ie, 2 influenza A and 2 influenza B strains) and safety data through Day 28. Data concerning secondary and exploratory endpoints will be included in the unblinded review of Days 0 and 28 as they become available. For the review, treatment codes will only be unblinded after the data are deemed ready for the analysis after all subjects have completed the Day 28 visit and the data are monitored. The determination of the readiness will be based on the blinded review of outstanding queries of critical data points. Given the time-consuming nature of the microneutralization, these data may be presented only in the final CSR or an addendum (see Section 10.6.2).

In order to execute this review, a select group of trial staff will be unblinded at the CRO and at Novavax. All personnel unblinded to the trial data will be documented. No individual unblinded at a subject treatment level will be involved in follow-up safety monitoring. Specifically, personnel at the clinical trial site including, investigators and trial staff, research site, immunology laboratory, and trial subjects will remain blinded to treatment assignments until the end of trial (ie, Day 364).

Since trial procedures and monitoring practices will not change following the review and the trial will not be terminated prematurely on the basis of these data, no decision cut points or stopping rules will be stipulated. Immunogenicity and safety analyses from the unblinded review may be presented in an abbreviated unblinded clinical study report (CSR) drafted by the Sponsor that may be submitted to regulatory authorities as needed.

# 10.6.2 Final Clinical Study Report

The final CSR will present the balance of all safety and immunogenicity (if any) data through Day 364 (the scheduled end of trial). The database will be locked and the final CSR prepared, when all of the above data have been entered, reviewed, and all queries related to the data have been addressed. Any decisions to deviate from the planned analyses will be described in detail in the final CSR.

# 10.7 Computer Methods

Statistical analyses will be performed using SAS® version 9.3 or greater under a Windows operating system.

#### 11 TRIAL LEGAL AND ETHICAL REQUIREMENTS

# 11.1 Compliance with Regulatory Requirements

This trial will be conducted in accordance with the protocol, the Declaration of Helsinki (amended Fortaleza, Brazil, 2013), International Conference on Harmonisation (ICH) GCP Guidelines, and the US FDA regulatory requirements.

### 11.2 Ethics Committee

This trial will be conducted under the auspices of a properly-constituted IRB, as defined by US regulatory requirements, and in accordance with the Declaration of Helsinki (amended Fortaleza, Brazil, 2013). This committee will review and approve all aspects of the trial, including the protocol and ICF to be used, any and all advertising or informational materials, and any modifications made to the protocol and ICF, prior to, or during the trial. Prior to initiation of clinical activity, investigators will provide Novavax with a copy of the communication from the IRB indicating approval of the protocol and ICF. In the event that a central IRB is used, Novavax will provide copies of correspondence to the investigators. All changes to the protocol or ICF must be reviewed and approved prior to implementation, except where necessary to eliminate apparent immediate hazards to human subjects.

If applicable, the investigators will be responsible for obtaining annual IRB renewal throughout the duration of the trial. Copies of the investigators' annual report to the IRB and copies of the IRB continuance of approval must be furnished to Novavax.

#### 11.3 Informed Consent

The investigators or designated site trial staff members will be responsible for obtaining written informed consent (and any applicable local or state regulatory documentation), signed and dated by each subject, prior to his/her participation in the trial. Informed consent will be obtained from a subject after a full explanation of the purpose of the trial, the risks and discomforts involved, potential benefits, etc, have been provided by the investigators, both verbally and in writing. The original signed copy of the ICF must be maintained in the institution's records and will be subject to inspection by a representative of Novavax and/or regulatory agencies. The subject will also be given a copy of the signed consent form.

# 11.4 Required Site Documentation

The following documents must be provided to Novavax or its designee prior to the start of the trial:

- Current *Curriculum Vitae* and medical licenses (as applicable) for the principal investigator and all sub-investigators,
- Financial Disclosure Forms from the principal investigator and all sub-investigators,
- Signed protocol and amendments (if any),

- Copy of correspondence from the IRB indicating approval of the protocol, ICF, and any site-specific trial advertisements, signed by the IRB chairperson or designee, and containing the name and address of the IRB,
- Membership roster of the IRB, listing names and occupations. If an investigator
  participating in this trial is an IRB member, documentation should be provided of his/her
  abstention from voting on this protocol,
- ICF reviewed and approved by the IRB, or a revised document if changes were requested by the committee with the IRB stamp and date, and
- Reference ranges for all safety tests required in the protocol and documentation of laboratory licensure if the trial site's local clinical laboratory will be used.

# 11.5 Subject Confidentiality

Individual subject medical information obtained as a result of this trial is considered confidential and disclosure to third parties, other than those cited below, is prohibited. Subject confidentiality will be further ensured by utilizing a subject identification code and subject initials. Relevant US national and local jurisdictions governing privacy rules and protection of human subjects will be followed in this trial.

In compliance with regulatory guidelines regarding the monitoring of clinical studies, and in fulfillment of the investigator's obligations to Novavax, it is required that data generated as a result of the trial be available for inspection, on request, by personnel from Novavax, CRO monitors representing Novavax, and/or regulatory agencies. These shall include all trial relevant documentation, including medical histories to verify eligibility, laboratory test results to verify transcription accuracy, treatment and diagnostic reports, and admission/discharge summaries for hospital admissions occurring while the subject is on-trial.

As part of the required content of the informed consent, subjects must be informed that their records will be reviewed by Novavax and/or regulatory agencies. Should access to the medical record require a separate waiver or authorization, it is the investigator's responsibility to obtain such permission from the subject in writing before the subject is entered into the trial.

### 11.6 Disclosure of Information

Information concerning the investigational Quad-NIV and patent application processes, scientific data, or other pertinent information is confidential and remains the property of Novavax. The investigator may use this information for the purposes of the trial only. It is understood by the investigator that Novavax will use information developed in this clinical trial in connection with the development of the investigational vaccine and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical trial, the investigator understands that he/she has an obligation to provide complete test results and all data developed during this trial to Novavax. Authorization to publish or otherwise publically disclose the results of this trial is strictly governed by the terms set forth in the clinical trial agreement.

### 12 REFERENCES

CDC. Estimates of Deaths Associated with Seasonal Influenza - United States, 1976-2007. MMWR Morb Mortal Wkly Rep (2010); 59(33): 1057-62.

CDC. (2017). Seasonal Influenza Vaccine Effectiveness, 2005-2017. Retrieved 19 April 2018 from <a href="https://www.cdc.gov/flu/vaccines-work/past-seasons-estimates.html">https://www.cdc.gov/flu/vaccines-work/past-seasons-estimates.html</a>.

CDC. (2019 -a). Influenza Vaccine - United States, 2018-19 Influenza Season. Retrieved 27 March 2019 from <a href="https://www.cdc.gov/flu/vaccines-work/past-seasons-estimates.html">https://www.cdc.gov/flu/vaccines-work/past-seasons-estimates.html</a>.

CDC. (2019 -b). What You Should Know and Do This Flu Season If You Are 65 Years and Older. Retrieved 27 March 2019, from <a href="https://www.cdc.gov/flu/highrisk/index.htm">https://www.cdc.gov/flu/highrisk/index.htm</a>.

Coffman RL, Sher A, Seder RA. Vaccine Adjuvants: Putting Innate Immunity to Work. Immunity (2010); 33(4): 492-503.

DiazGranados CA, Dunning AJ, Kimmel M, et al. Efficacy of High-Dose Versus Standard-Dose Influenza Vaccine in Older Adults. N Engl J Med (2014); 371(7): 635-45.

Doyle JD, Chung JR, Kim SS, et al. Interim Estimates of 2018-2019 Seasonal Influenza Vaccine Effectiveness - United States, February 2019. MMWR Morb Mortal Wkly Rep (2019); 68(6): 135-9.

FDA. (2019). Vaccines Licensed for Use in the United States. Retrieved 27 March 2019, from https://www.fda.gov/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM093833.

Flannery B, Chung J, Belongia EA, et al. (2018). Interim Estimates of 2017-18 Seasonal Influenza Vaccine Effectiveness - United States, February 2018. MMWR Morb Mortal Wkly Rep (2018); 67(6): 180-5.

Griffin MR, Monto AS, Belongia EA, et al. Effectiveness of Non-Adjuvanted Pandemic Influenza A Vaccines for Preventing Pandemic Influenza Acute Respiratory Illness Visits in 4 U.S. Communities. PLoS One (2011); 6(8): e23085.

Grohskopf LA, Sokolow LZ, Broder KR, et al. Prevention and Control of Seasonal Influenza with Vaccines. MMWR Recomm Rep (2016); 65(5): 1-54.

McLean HQ, Thompson MG, Sundaram ME, et al. Influenza Vaccine Effectiveness in the United States During 2012-2013: Variable Protection by Age and Virus Type. J Infect Dis (2015); 211(10): 1529-40.

Monto AS. Moving Toward Improved Influenza Vaccines. J Infect Dis (2017); 215(4): 500-2.

Mullooly JP, Bridges CB, Thompson WW, et al. Influenza- and RSV-Associated Hospitalizations Among Adults. Vaccine (2007); 25(5): 846-55.

Ohmit SE, Thompson MG, Petrie JG, et al. Influenza Vaccine Effectiveness in the 2011-2012 Season: Protection Against Each Circulating Virus and the Effect of Prior Vaccination on Estimates. Clin Infect Dis (2014); 58(3): 319-27.

Paules C and Subbarao K. Influenza. Lancet (2017); 390(10095): 697-708.

Reed C, Kim IK, Singleton JA, et al. Estimated Influenza Illnesses and Hospitalizations Averted by Vaccination - United States, 2013-14 Influenza Season. MMWR Morb Mortal Wkly Rep (2014); 63(49): 1151-4.

Reed C, Chaves SS, Daily Kirley P, et al. Estimating Influenza Disease Burden from Population-Based Surveillance Data in the United States. PLoS One (2015); 10(3): e0118369.

Shinde V, Fries L, Wu Y, et al. Improved Titers Against Influenza Drift Variants with a Nanoparticle Vaccine. N Engl J Med (2018); 378(24): 2346-8.

Skowronski DM, Chamber C, Sabaiduc S, et al. A Perfect Storm: Impact of Genomic Variation and Serial Vaccination on Low Influenza Vaccine Effectiveness During the 2014-2015 Season. Clin Infect Dis 2016; 63(1): 21–32.

Smith G, Liu Y, Flyer D, et al. Novel Hemagglutinin Nanoparticle Influenza Vaccine with Matrix-M<sup>TM</sup> Adjuvant Induces Hemagglutination Inhibition, Neutralizing, and Protective Responses in Ferrets Against Homologous and Drifted A(H3N2) Subtypes. Vaccine 2017; 35(40): 5366-72.

Sullivan SG, Chilver MB, Carville KS, et al. Low Interim Influenza Effectiveness, Australia, 1 May to 24 September 2017. Euro Surveill (2017); 22(43): 10.2807/1560-7917.

Treanor JJ, Talbot HK, Ohmit SE, et al. Effectiveness of Seasonal Influenza Vaccines in the United States During a Season with Circulation of All Three Vaccine Strains. Clin Infect Dis (2012); 55(7): 951-9.

VRBPAC. (2018). Summary Minutes: 151<sup>st</sup> Vaccines and Related Biological Products Advisory Committee. Retrieved 29 March 2018. https://www.fda.gov/downloads/AdvisoryCommittees/CommitteesMeetingMaterials/BloodVaccinesandOtherBiologics/VaccinesandRelatedBiologicalProductsAdvisoryCommittee/UCM602610.pdf.

VRBPAC. (2019). Summary Minutes: 152<sup>nd</sup> Vaccines and Related Biological Products Advisory Committee. Retrieved 27 March 2019. https://www.fda.gov/downloads/AdvisoryCommittees/CommitteesMeetingMaterials/BloodVaccinesandOtherBiologics/VaccinesandRelatedBiologicalProductsAdvisoryCommittee/UCM6 33766.pdf.

WHO (2011). Manual for the Laboratory Diagnosis and Virological Surveillance of Influenza. WHO Global Influenza Surveillance Network. Retrieved 18 October 2017, from http://whqlibdoc.who.int/publications/2011/9789241548090\_eng.pdf.

WHO. (2017). Recommended Composition of Influenza Virus Vaccines for Use in the 2017-2018 Northern Hemisphere Influenza Season. Retrieved 18 October 2017, from https://www.who.int/influenza/vaccines/virus/recommendations/2017\_18\_north/en/.

WHO. (2018). Recommended Composition of Influenza Virus Vaccines for Use in the 2018-2019 Northern Hemisphere Influenza Season. Retrieved 29 March 2018, from https://www.who.int/influenza/vaccines/virus/recommendations/2018\_19\_north/en/.

WHO. (2019). Recommended Composition of Influenza Virus Vaccines for Use in the 2019-2020 Northern Hemisphere Influenza Season. Retrieved 27 March 2019, from https://www.who.int/influenza/vaccines/virus/recommendations/2019\_20\_north/en/.

Zimmerman RK, Nowalk MP, Chung J, et al. 2014-2015 Influenza Vaccine Effectiveness in the United States by Vaccine Type. Clin Infect Dis (2016); 63(12): 1564-73.

Zost SJ, Parkhouse K, Gumina ME, et al. Contemporary H3N2 Influenza Viruses Have a Glycosylation Site that Alters Binding of Antibodies Elicited by Egg-Adapted Vaccine Strains. Proc Natl Acad Sci U S A (2017); 114(47): 12578-83.

# APPENDIX 1 - QNIV-E-301 TRIAL PROCEDURES SCHEDULE

| Trial Day: | 0 | 3 | 7 | 28 | 90 | 182 | 364 |
|---|---|---|---|---|---|---|---|
| Window (days): | | ± 1 | ± 1 | ± 4 | ± 7 | ± 7 | ± 14 |
| <b>Trial Procedures</b> | | | | | | | |
| Trial Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical/Medication History | X | | | | | | |
| Physical Exam | X | | X [4] | X [4] | | X [4] | |
| Vital Signs | X [1] | | X | X | | X | |
| Serology | X | | | X | | X | |
| PMBC for CMI | $X^{[5]}$ | | $X^{[5]}$ | $X^{[5]}$ | | $X^{[5]}$ | |
| Trial Treatment Injection | X | | | | | | |
| Adverse Event Review [2] | X | X | X | X | X | X | X |
| Concomitant Medications<br>Review [2] | X | X | X | X | X | X | X |
| Subject Diary Review | | | | X [3] | | | |
| End of Trial | | | | | | | X |

Note: Procedures shaded in grey are performed via scripted telephone call.

<sup>[1]</sup> Vital signs to be captured pre-vaccination and between 30 to 60 minutes post-vaccination.

<sup>[2]</sup> All adverse events and concomitant medications taken will be collected through Day 28; thereafter, only MAEs, SAEs, and SNMCs and medications taken for these events will be collected.

<sup>[3]</sup> The subject diary will be reviewed by the investigator and collected at the Day 28 visit.

<sup>[4]</sup> If needed, a physical examination may be performed, based on the investigator's discretion.

<sup>[5]</sup> To be collected from a subset of approximately 140 subjects from several pre-designated clinical sites.

# APPENDIX 2 - QNIV-E-301 SUBJECT DIARY CARD (DRAFT)

| Subject ID Subject Initials | | | | | | | | | /- | | | - 1 | | | | | | | - 77 | | | | - | | | - 2 | | "" GRADING FOR DIARRHEA 0 = Normal | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| JS | Day | of Va<br>(Da | | lon | Day 1 | | Day 1 | | | | Day 1 | | | | Day 1 | | | Day 2 | | | Day 3 | | | Day 4 | | | Day 5 | | Day 6 | Ongoing after Day 67 | No noticeable symptom<br>1 = Mild |
| | Date: | | | | Date | | | | Date: | | | | Date: | | | Date | | | 0 | Date: | | | Date: | | | | | 1 to 3 unformed (loose) stools<br>within a 24-hour period | | | |
| | | | _/ | | - | / | 1 | | | | <i></i> | | | | | 4 | // | | | | _/ | | | | | - | | 2 = Moderate<br>4 to 5 unformed (loose) stools | | | |
| ORAL TEMPERATURE | | | T | | | | F | | | | F | | | | *F | | | F | | | F | | | | _TF | | (tick the box if<br>symptom is still continuing<br>after Day 6) | within a 24-hour period 3 = Severe 6 or more loose stools within a 24-hour period, | | | |
| | | NO SY | YMPT | DMS | 0 | NO S | YMPTO | OMS | ۵ | NO SY | мртом | 5 | □ NO SYMPTOMS | | | 0 | □ NO SYMPTOMS | | | □ NO SYMPTOMS | | | 0 | NO SYI | APTON | AS | | or requires intravenous hydration *** GRADING FOR NAUSEA AND VOMITING | | | |
| GENERAL SYMPTOMS | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 3 | 0 | 1 | 2 | | 0 1 | 2 | 3 | 0 | î | 2 | 3 | | 0 = Normal No noticeable symptom 1 = Mild | | | |
| Chills | | T | | | | | | | | | | | | | | | | | | | | | | | | | 0 | No interference with activity or<br>1 to 2 episodes within a 24-hour period | | | |
| Muscle Pain | | - | | - 1 | | | | | | | -1 | | | | | | | | - 4 | | | | | - | | - 6 | 0 | 2 = Moderate<br>Some interference with activity or | | | |
| ioint Pain | | | | - 2 | | | | | | | - 1 | | | - | | | | | 1 | | | 7 | | | _ | 7 | 0 | >2 episodes within a 24-hour period<br>3 = Severe | | | |
| Diarrhea | | | | - 8 | | | | - | | | 1 | | | | | | | | | | | | | | | - 19 | | Prevents daily activity or requires | | | |
| Nausea *** | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | intravenous hydration O = NORMAL | | | |
| Vomiting *** | | | | | | | | | | | | | | | | | | | | | | | | | | | | No noticeable symptom or finding | | | |
| Headache | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | 1 = MILD | | | |
| Fatigue | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | <ul> <li>Noticeable discomfort/pain, or symptom<br/>that does not interfere with activities of</li> </ul> | | | |
| RESPIRATORY/FACIAL SYMPTOMS | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 3 | 0 | 1 | 2 | | 0 1 | 2 | 3 | 0 | 1 | 2 | 3 | | daily living 2 = MODERATE | | | |
| Cough | | _ | | | | | | | | | | | | | | | | | | | | | | | | | 0 | Moderate discomfort/pain, or symptom that limits but does not stop activities of daily living 3 = SEVERE Sewere pain of symptoms that stop activities of daily living and may require medical treatment | | | |
| Difficulty Breathing | | | | - 2 | | | | | | | -1 | | | | | | | | - | | | | | | | - 6 | | | | | |
| Chest Tightness | | | | - 2 | | | | | | | | | | == | | | | | 4 | | | | | | _ | - 1 | 0 | | | | |
| Wheezing | | | | | | | | | | | 1 | | | | | | | | | | | | | | | | | | | | |
| Sore Throat | | | | | | | | | | | Ī | | | | | | | | | | | | | | | | 0 | | | | |
| Difficulty Swallowing | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | | | | |
| Hoarseness | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | | | | |
| Eye Redness | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | | | | |
| Eyelid Swelling | | H | | - 3 | | | | | | | - 1 | | | | | | | | - | | | | | | | - 7 | | | | | |
| Factal Swelling | | | | - 2 | | | | | | | | | | | | | | | 1 | | | | | | - | - 1 | 0 | d . | | | |
| INJECTION SITE SYMPTOMS | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 3 | 0 | 1 | 2 | 8 | 0 1 | 2 | 3 | 0 | 1 | 2 | 3 | | O = NORMAL | | | |
| Pain | | | | | | | | | | | | | - 10 | 20 | | | | | 2 | | | | | | | - 0 | 0 | No noticeable symptom 1 = MILD | | | |
| Bruising* | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | Noticeable discomfort or tenderness | | | |
| Redness* | | | | | | | | | | | | | | | | | | | | | | | | | | | | that does not interfere will normal activit 2 = MODERATE | | | |
| Swelling* | | | | | | | | | | | | | | | | | | | | | | | | | | | 0 | Moderate discomfort or tenderness that | | | |
| Please complete the questions below by cho<br>Any box marked with a "YES" will require ac | oosing | either<br>al info | "Yes" | or "No | o." Circ | de you | r respo | nse. | | | | | | | | | | | | | | | | | | | | <ul> <li>casuses some limitation of normal activi</li> <li>3 = SEVERE Severe pain at rest, immobilizes the </li> </ul> | | | |
| Have your medications changed or are you taking any new medications? | Y | s | | NO | , | res | 110 | NO | YE | s | NO | | YES | | NO: | , | 'ES | NO | | YES | | NO. | YE | s | NC | ) | | injected arm and prevents normal daily<br>activity *SEE SUBJECT MEASUREMENT TOOL | | | |
| If yes, please record in the Medication Log. Did you visit a doctor? | | | | | | | | | | | | | | | | | | | | | | | | | | | | INSTRUCTIONS | | | |
| if yes, please record the reason for seeking<br>medical attention in the Doctor Visit Log. | YI | S | - 1 | NO | , | rES | , | NO | YE | s | NO | | YES | | NO | , | 'ES | NO | | YES | , | NO. | YE | S | NC | ) | | | | | |
| Did you have any other symptoms?<br>If yes, please list them in the "Other<br>Symptoms Log" on page 8. | Y | S | 1 | NO | Ŋ | /ES | 1 | NO. | YE | s | NO | | YES | | NO: | Ŋ | 'ES | NO | | YES | | NO. | YE | s | NO | ) | | | | | |

<sup>\*</sup>A subject diary will be provided to all subjects to record solicited and unsolicited adverse events experienced, concomitant medications used, and any medical visits/procedures sought, within the first 7 days following the Day 0 vaccination. The above is a sample excerpt from such a diary. It is provided for informational purposes only and may differ from the actual diary issued to subjects.

# **APPENDIX 3 - QNIV-E-301 BLOOD DRAW SCHEDULE**

| Trial Visit Day | Amount of Blood Drawn for<br>Immunogenicity Assessment (mL) | Amount of Blood Drawn for<br>CMI Assessment (mL) |
|---|---|---|
| Day 0 (pre-vaccination) | 20 | 27 <sup>[1]</sup> |
| Day 7 ( $\pm 1 day$ ) | | 27 <sup>[1]</sup> |
| Day 28 (±4 days) | 20 | 27 <sup>[1]</sup> |
| Day 182 (±7 days) | 20 | 27 <sup>[1]</sup> |
| TOTAL FOR ENTIRE<br>TRIAL (mL) | 60 – 16 | 8 [2] |

<sup>[1]</sup> To be collected from a subset of approximately 140 subjects from several pre-designated clinical sites.

<sup>[2]</sup> Most subjects will provide up to 60 mL of blood in the trial. A subset of approximately 140 subjects from several pre-designated clinical sites will provide up to 168 mL.

#### APPENDIX 4 – QNIV-E-301 SUBJECT MEASUREMENT TOOL

(Do not use this page in clinic, as it may not be to exact scale)



The Subject Measurement Tool consists of a transparent set of concentric circles with diameters that correspond to the ranges in the toxicity grading scale (2.5, 5, and 10 cm, in diameter). Subjects are instructed to overlay the template over the injection site for any reaction that can be visually observed (eg, redness, swelling, bruising). An assessment of severity is then made by determining the circle that best describes the size of the reaction: reactions that are smaller than Circle A (2.5 cm) are considered Grade 0; reactions larger than Circle A but equal to or smaller than Circle B (5 cm) are considered Grade 1; reactions larger than Circle B but equal to or smaller than Circle C (10 cm) are considered Grade 2; reactions larger than Circle C are considered Grade 3. The table below summarizes the severity grading for visible injection site reactions based on size.

**Definition of Severity Grading for Visible Local Adverse Events** 

| Severity Grade | Injection Site Grading Description |
|---|---|
| 0 - Normal | Reaction size fits inside Circle A |
| 1 - Mild | Reaction size larger than Circle A, but fits inside Circle B |
| 2 - Moderate | Reaction size larger than Circle B, but fits inside Circle C |
| 3 - Severe | Reaction size larger than Circle C |